CLINICAL TRIAL: NCT03803202
Title: A Phase 1/2, Randomized, Single Ascending Dose Study in Adults (Stage 1) and Randomized, Single Ascending Dose-Finding Study (Stage 2) in Elderly Subjects With ASP3772, a Pneumococcal Vaccine
Brief Title: A Single Ascending Dose Study in Adults (Stage 1) and Single Ascending Dose-Finding Study (Stage 2) in Elderly Subjects With ASP3772, A Pneumococcal Vaccine
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Affinivax, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: 219659; 3772-CL-1001 (Other: Affinivax Inc. Study ID)
Record Dates: First submitted 2019-01-11; First posted 2019-01-14 (Actual); Results first posted 2023-12-21 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-11

CONDITIONS: Pneumonia, Bacterial; Healthy Volunteers; Pneumococcal Disease
Keywords: Pneumococcal vaccine; Vaccine; Pneumococccal Disease; ASP3772
MeSH Terms: conditions — Pneumonia, Bacterial; Pneumococcal Infections | interventions — 13-valent pneumococcal vaccine; 23-valent pneumococcal capsular polysaccharide vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Stage 1, Group 1 Adults, ASP3772 Low dose (Experimental): Healthy adults aged 18 to 64 years received a low dose [1 microgram (μg)] of ASP3772 intramuscularly on Day 1.
  Interventions: Biological: ASP3772
- Stage 1, Group 1 Adults, ASP3772 Medium dose (Experimental): Healthy adults aged 18 to 64 years received a medium dose (2 μg) of ASP3772 intramuscularly on Day 1.
  Interventions: Biological: ASP3772
- Stage 1, Group 1 Adults, ASP3772 High dose (Experimental): Healthy adults aged 18 to 64 years received a high dose (5 μg) of ASP3772 intramuscularly on Day 1.
  Interventions: Biological: ASP3772
- Stage 1, Group 1, PCV13 Pooled Comparator (Active Comparator): Healthy adults aged 18 to 64 years received a single dose of PCV13 0.5 milliliter (mL) intramuscularly on Day 1. Data from participants in each group given PCV13 were pooled for comparison with each ASP3772 dose group (ASP3772 low dose, ASP3772 medium dose and ASP3772 high dose).
  Interventions: Biological: PCV13
- Stage 2, Group 2 Older Adults, ASP3772 Low dose (Experimental): Healthy older adults aged 65 to 85 years received a low dose (1 μg) of ASP3772 intramuscularly on Day 1.
  Interventions: Biological: ASP3772
- Stage 2, Group 2 Older Adults, ASP3772 Medium dose (Experimental): Healthy older adults aged 65 to 85 years received a medium dose (2 μg) of ASP3772 intramuscularly on Day 1.
  Interventions: Biological: ASP3772
- Stage 2, Group 2 Older Adults, ASP3772 High dose (Experimental): Healthy older adults aged 65 to 85 years received a high dose (5 μg) of ASP3772 intramuscularly on Day 1.
  Interventions: Biological: ASP3772
- Stage 2, Group 2, PCV13 Pooled Comparator (Active Comparator): Older adults aged 65 to 85 years received a single dose of PCV13 0.5 mL intramuscularly on Day 1. Data from participants in each group given PCV13 were pooled for comparison with each ASP3772 dose group (ASP3772 low dose, ASP3772 medium dose and ASP3772 high dose).
  Interventions: Biological: PCV13
- Stage 2, Group 3, PPSV23 Comparator (Active Comparator): Older adults aged 65 to 85 years who had been previously vaccinated with PCV13, were enrolled and received a single of dose PPSV23 on Day 1.
  Interventions: Biological: PPSV23

INTERVENTIONS:
Biological: ASP3772 — Participants received a single dose of ASP3772 (ASP3772 low dose, ASP3772 medium dose and ASP3772 high dose) intramuscularly
  Arms: Stage 1, Group 1 Adults, ASP3772 High dose; Stage 1, Group 1 Adults, ASP3772 Low dose; Stage 1, Group 1 Adults, ASP3772 Medium dose; Stage 2, Group 2 Older Adults, ASP3772 High dose; Stage 2, Group 2 Older Adults, ASP3772 Low dose; Stage 2, Group 2 Older Adults, ASP3772 Medium dose
Biological: PCV13 — Participants received a single dose of PCV13 intramuscularly.
  Other Names: Prevnar 13
  Arms: Stage 1, Group 1, PCV13 Pooled Comparator; Stage 2, Group 2, PCV13 Pooled Comparator
Biological: PPSV23 — Participants received a single dose of PPSV23 intramuscularly.
  Other Names: Pneumovax 23
  Arms: Stage 2, Group 3, PPSV23 Comparator

SUMMARY:
The purpose of the study is to evaluate the safety, tolerability, and immunogenicity of 3 different dose levels of ASP3772 in comparison to the active comparator Prevnar 13® (PCV13) in adults 18 to 64 years of age in Stage 1. Stage 2 will evaluate the safety, tolerability, and immunogenicity of 3 different dose levels of ASP3772 in comparison to the active comparator PCV13 in elderly 65 to 85 years of age. In addition, Stage 2 will evaluate the immunogenicity of 3 different dose levels of ASP3772 relative to the response seen following administration of Pneumovax® 23 (PPSV23) for the serotypes not included in PCV13.

DETAILED DESCRIPTION:
The study population will consist of 3 different groups: Group 1 - Stage 1 PCV13 naïve participants randomized within 3 sequential cohorts to ASP3772 or PCV13; Group 2 - Stage 2 PCV13 naïve participants randomized within 3 sequential cohorts to ASP3772 or PCV13; and Group 3 - Stage 2 participants previously vaccinated with PCV13 that will receive PPSV23.

ELIGIBILITY:
Inclusion Criteria:

* Stage 1: Subject is healthy male or female between 18 and 64 year of age inclusive, at screening.
* Stage 2: Subject is a male or female between 65 and 85 years of age, inclusive, at screening who is healthy or has chronic controlled, stable disease with no change in disease severity, medical therapy and no hospitalization records in last 12 weeks as determined by medical history, physical examination and laboratory data.
* A female subject is eligible to participate if not pregnant and at least 1 of the following conditions applies:

  * Not a woman of childbearing potential (WOCBP) OR
  * WOCBP who agrees to follow the contraceptive guidance at screening and for at least 28 days after the study vaccine administration.
* Female subject must agree not to breastfeed starting at screening and for 28 days after the study vaccine administration.
* Female subject must not donate ova starting at screening and for 28 days after the study vaccine administration.
* A male subject with female partner(s) of childbearing potential must agree to use contraception at screening and for at least 28 days after the study vaccine administration.
* Male subject must not donate sperm starting at screening and for 90 days after the study vaccine administration.
* Male subject with a pregnant or breastfeeding partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy or time partner is breastfeeding at screening and for 28 after the study vaccine administration.
* Subject agrees not to participate in another interventional study while participating in the present study.

Exclusion Criteria:

* Subject has a known or suspected hypersensitivity to ASP3772, its comparators or any components of the formulations used.
* Subject has had previous exposure with ASP3772.
* Subject has had known previous exposure with PPSV23.
* Subject has received PCV13 or any other licensed or investigational pneumococcal vaccine at any time. (Note: This exclusion criterion is not applicable to Group 3; those subjects 65 to 85 years of age who previously received immunization with PCV13. Prior PCV13 immunization should have taken place no less than 10 months and no more than 2 years prior to study vaccine administration. These subjects are eligible to be enrolled in the nonrandomized arm of Stage 2, Group 3.
* Subject has a history of microbiologically-proven invasive disease caused by S. pneumoniae.
* Subject has an immune disorder(s) (including autoimmune disease) and/or clinical conditions requiring immunosuppressive drugs.
* Subject has any evidence of any unstable or active clinically significant cardiovascular, gastrointestinal, endocrine, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal and/or other major disease or malignancy, e.g., uncontrolled hypertension, uncontrolled diabetes, heart failure, uncontrolled chronic obstructive pulmonary disease, end-stage renal disease.
* Subject has history of illicit drug(s) or alcohol abuse that will interfere with the protocol requirements and/or a positive urine drug test (for Stage 1 subjects only) at screening.
* Subject has any clinically significant history of allergic conditions including drug allergies, asthma or anaphylactic reactions, but excluding untreated asymptomatic seasonal allergies prior to study vaccine administration.
* Subject has a coagulation disorder contraindicating intramuscular immunization.
* Subject has a positive serology test for hepatitis B surface antigen (HBsAg), hepatitis A virus antibodies (immunoglobulin M), hepatitis C virus antibodies (anti-HCV) confirmed by reflex testing (HCV-RNA) or antibodies to human immunodeficiency virus (HIV) type 1 and/or type 2 at screening.
* Subject has/had febrile illness (> 100.4°F oral equivalent) or symptomatic, viral, bacterial (including upper respiratory infection) or fungal (noncutaneous) infection within 1 week prior to day 1.
* Subject has any clinically significant abnormality from the physical examination, ECG and clinical laboratory tests during screening.
* Subject is unlikely to adhere to study procedures, keep appointments, is planning to relocate during the study or cannot be adequately followed for safety according to the protocol.
* Subject has any other condition, which precludes the subject's participation in the study.
* Subject has received any vaccines within 30 days prior of receipt of the study vaccine (exception: Influenza virus vaccine given according to recommended guidelines must be given at least 7 days prior to receiving study vaccine).
* Subject has had significant blood loss, donated 1 unit (450 mL or more) or received transfusion of any blood or blood products within 60 days or donated plasma within 7 days prior to day 1.
* Subject has received any systemically absorbed antibiotics during the 7-day period prior to day 1.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 630 (Actual)
Dates: Start 2019-01-24 (Actual); Primary Completion 2020-09-28 (Actual); Study Completion 2020-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (25):
- United States (25):
  - Advanced Clinical Research-Rancho Paseo, Banning, California
  - Artemis Institute, San Diego, California
  - Artemis Institute, San Marcos, California
  - Research Centers of America, Hollywood, Florida
  - Meridian Clinical Research, Savannah, Georgia
  - Sundance Clinical Research, St Louis, Missouri
  - Meridian Clinical Research, Norfolk, Nebraska
  - United Medical Associates, Binghamton, New York
  - PMG Research of Raleigh, Raleigh, North Carolina
  - PMG Research of Hickory, LLC, Rocky Mount, North Carolina
  - Piedmont HealthCare, PA, Statesville, North Carolina
  - Wilmington Health, Wilmington, North Carolina
  - PMG Research of Winston-Salem, LLC, Winston-Salem, North Carolina
  - Tekton Research - George Town, Yukon, Oklahoma
  - PMG Research, Knoxville, Tennessee
  - Advanced Clinical Research Institute, Cedar Park, Texas
  - Texas Healthcare, PLLC, Fort Worth, Texas
  - Benchmark Research, Fort Worth, Texas
  - Texas Center for Drug Development, Houston, Texas
  - Healthcare Associatiates of Texas, McKinney, Texas
  - DM Clinical Research, Pearland, Texas
  - Benchmark Research, San Angelo, Texas
  - Clinical Trials of Texas, San Antonio, Texas
  - Martin Diagnostic Clinic, Tomball, Texas
  - CRA of Tidewater Inc, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as compounds terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Conditions and exceptions are described under the Sponsor Specific Details for Astellas on www.clinicalstudydatarequest.com.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicalstudydatarequest.com/

REFERENCES:
- [Derived] Borys D, Rupp R, Smulders R, Chichili GR, Kovanda LL, Santos V, Malinoski F, Siber G, Malley R, Sebastian S. Safety, tolerability and immunogenicity of a novel 24-valent pneumococcal vaccine in toddlers: A phase 1 randomized controlled trial. Vaccine. 2024 Apr 11;42(10):2560-2571. doi: 10.1016/j.vaccine.2024.02.001. Epub 2024 Feb 14. PMID 38360475
- [Derived] Chichili GR, Smulders R, Santos V, Cywin B, Kovanda L, Van Sant C, Malinoski F, Sebastian S, Siber G, Malley R. Phase 1/2 study of a novel 24-valent pneumococcal vaccine in healthy adults aged 18 to 64 years and in older adults aged 65 to 85 years. Vaccine. 2022 Jul 29;40(31):4190-4198. doi: 10.1016/j.vaccine.2022.05.079. Epub 2022 Jun 9. PMID 35690500

RESULTS

PARTICIPANT FLOW:
Recruitment Details: For Stage 1 out Of the 178 participants who provided informed consent only 127 participants were enrolled and randomized into the study.
  For Stage 2 Group 2 and Stage 2 Group 3 - out of 757 participants, A total of 390 participants were enrolled and randomized to Group 2 and 113 participants were enrolled in Group 3.
Pre-assignment Details: Analysis of this study results were reported for the PSV13 Pooled Comparator group to compare with the ASP3772 groups. According to the pre-specified analysis plan, data collected for participant flow, baseline characteristics, Outcome Measures and adverse events reporting were not analyzed for the individual PCV13 groups.
Groups:
- Stage 2, Group 2 Older Adults, ASP3772 High Dose: Healthy older adults aged 65 to 85 years, received a high dose (5 μg) of ASP3772 intramuscularly on Day 1.
- Stage 2, Group 3, PPSV23 Comparator: Older adults aged 65 to 85 years, who had been previously vaccinated with PCV13, were enrolled and received a single of dose PPSV23 on Day 1.
Period: Overall Study
Arm/Group | Stage 1, Group 1 Adults, ASP3772 Low Dose | Stage 1, Group 1 Adults, ASP3772 Medium Dose | Stage 1, Group 1 Adults, ASP3772 High Dose | Stage 1, Group 1, PCV13 Pooled Comparator | Stage 2, Group 2 Older Adults, ASP3772 Low Dose | Stage 2, Group 2 Older Adults, ASP3772 Medium Dose | Stage 2, Group 2 Older Adults, ASP3772 High Dose | Stage 2, Group 2, PCV13 Pooled Comparator | Stage 2, Group 3, PPSV23 Comparator
Started (Started = All enrolled participants) | 30 | 32 | 32 | 33 | 100 | 107 | 86 | 97 | 113
Vaccinated (Vaccinated = number of participants who completed the vaccination) | 30 | 31 | 32 | 33 | 100 | 107 | 86 | 97 | 113
Completed | 30 | 31 | 31 | 32 | 99 | 106 | 85 | 96 | 113
Not Completed | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0
Not completed — Other | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Stage 1, Group 1 Adults, ASP3772 Low Dose: Healthy adults aged 18 to 64 years received a low dose (1 μg) of ASP3772 intramuscularly on Day 1.
- Stage 1, Group 1, PCV13 Pooled Comparator: Healthy adults aged 18 to 64 years received a single dose of PCV13 0.5 mL intramuscularly on Day 1. Data from participants in each group given PCV13 were pooled for comparison with each ASP3772 dose group (ASP3772 low dose, ASP3772 medium dose and ASP3772 high dose).
- Total: Total of all reporting groups
Arm/Group | Stage 1, Group 1 Adults, ASP3772 Low Dose | Stage 1, Group 1 Adults, ASP3772 Medium Dose | Stage 1, Group 1 Adults, ASP3772 High Dose | Stage 1, Group 1, PCV13 Pooled Comparator | Stage 2, Group 2 Older Adults, ASP3772 Low Dose | Stage 2, Group 2 Older Adults, ASP3772 Medium Dose | Stage 2, Group 2 Older Adults, ASP3772 High Dose | Stage 2, Group 2, PCV13 Pooled Comparator | Stage 2, Group 3, PPSV23 Comparator | Total
Number analyzed (Participants) | 30 | 32 | 32 | 33 | 100 | 107 | 86 | 97 | 113 | 630
Age, Customized [Count of Participants; unit: Participants]
  >=18 to <65 years | 30 | 32 | 32 | 33 | 0 | 0 | 0 | 0 | 0 | 127
  >=65 to <75 years | 0 | 0 | 0 | 0 | 90 | 89 | 78 | 84 | 108 | 449
  >=75 to <=85 years | 0 | 0 | 0 | 0 | 10 | 18 | 8 | 13 | 5 | 54
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 21 | 21 | 23 | 64 | 55 | 44 | 52 | 70 | 369
  Male | 11 | 11 | 11 | 10 | 36 | 52 | 42 | 45 | 43 | 261
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 25 | 26 | 29 | 28 | 89 | 92 | 79 | 78 | 104 | 550
  Black or African American | 4 | 5 | 2 | 5 | 10 | 15 | 7 | 16 | 7 | 71
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 3
  Other | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), [Stage 1, Group 1]
Description: An AE is any untoward medical occurrence in a participant administered a study vaccine, and which does not necessarily have to have a causal relationship with this vaccination. A TEAE is defined as any AE with onset within 30 days from study vaccine administration. Medically attended TEAEs (MAAEs) are AEs for which the participant has received medical attention by medical personnel, or in an emergency room, or which led to hospitalization.
  A new-onset chronic disease TEAEs (NOCD) is defined as a MAAE which a) was absent at baseline; b) has not resolved at the follow-up telephone call; c) requires continuous medical care or attention. Potentially Immune Mediated medical condition TEAEs (PIMMCs) are defined as any AEs of autoimmune or auto inflammatory nature.
Time Frame: From Day 1, Up to Day 180
Population: The analysis was performed on the Safety Analysis Set (SAF) which consisted of all randomized participants who received a vaccination in this study with either ASP3772 or PCV13.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1, Group 1 Adults, ASP3772 Low Dose | Stage 1, Group 1 Adults, ASP3772 Medium Dose | Stage 1, Group 1 Adults, ASP3772 High Dose | Stage 1, Group 1, PCV13 Pooled Comparator
Number analyzed (Participants) | 30 | 31 | 32 | 33
Participants
  TEAE | 11 | 5 | 5 | 5
  Vaccine-Related TEAEs | 2 | 1 | 1 | 0
  Medically Attended TEAE | 3 | 3 | 0 | 1
  Potentially Immune Mediated TEAEs | 0 | 0 | 0 | 0
  NOCDs | 0 | 0 | 0 | 0
  Serious TEAEs | 0 | 0 | 0 | 0
  Serious Vaccine-Related TEAE | 0 | 0 | 0 | 0
  Death | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With TEAEs, [Stage 2, Group 2]
Description: An AE is any untoward medical occurrence in a participant administered a study vaccine, and which does not necessarily have to have a causal relationship with this vaccination. A TEAE is defined as any AE with onset within 30 days from study vaccine administration. Medically attended TEAEs (MAAEs) are AEs for which the participant has received medical attention by medical personnel, or in an emergency room, or which led to hospitalization.
  A new-onset chronic disease TEAEs (NOCD) is defined as a MAAE which a) was absent at baseline; b) has not resolved at the follow-up telephone call; c) requires continuous medical care or attention. Potentially Immune Mediated medical condition TEAEs (PIMMCs) are defined as any AEs of autoimmune or auto inflammatory nature. As specified in protocol, data was planned to be analyzed for PCV13 pooled comparator from each group given PCV13 to compare with each ASP3772 dose.
Time Frame: From Day 1, Up to Day 180
Population: The analysis was performed on the Safety Analysis Set which consisted of all randomized participants who received a vaccination in this study with either ASP3772 or PCV13.
Measure: Count of Participants; unit: Participants
Groups:
- Stage 2, Group 2 Older Adults, ASP3772 Low Dose: Healthy older adults aged 65 to 85 years, received a low dose (1 μg) of ASP3772 intramuscularly on Day 1.
- Stage 2, Group 2 Older Adults, ASP3772 Medium Dose: Healthy older adults aged 65 to 85 years, received a medium dose (2 μg) of ASP3772 intramuscularly on Day 1.
Arm/Group | Stage 2, Group 2 Older Adults, ASP3772 Low Dose | Stage 2, Group 2 Older Adults, ASP3772 Medium Dose | Stage 2, Group 2 Older Adults, ASP3772 High Dose | Stage 2, Group 2, PCV13 Pooled Comparator
Number analyzed (Participants) | 100 | 107 | 86 | 97
Participants
  TEAE | 25 | 26 | 28 | 14
  Vaccine-Related TEAEs | 5 | 5 | 8 | 3
  Medically Attended TEAE | 7 | 9 | 7 | 3
  New Onset Chronic TEAEs | 2 | 1 | 1 | 1
  Potentially Immune Mediated TEAEs | 0 | 0 | 0 | 0
  Serious TEAEs | 4 | 5 | 1 | 0
  Serious Vaccine-Related TEAE | 0 | 0 | 0 | 0
  Death | 0 | 1 | 0 | 0

3. Primary Outcome: Number of Participants With TEAEs, [Stage 2, Group 3]
Description: as for outcome 1
Time Frame: From Day 1, Up to Day 30
Population: The analysis was performed on the Safety Analysis Set which consisted of all randomized participants who received a vaccination in this study with PPSV23.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2, Group 3, PPSV23 Comparator
Number analyzed (Participants) | 113
Participants
  TEAE | 12
  Vaccine-Related TEAEs | 2
  Medically Attended TEAE | 1
  New Onset Chronic TEAEs | 0
  Potentially Immune Mediated TEAEs | 0
  Serious TEAEs | 0
  Serious Vaccine-Related TEAE | 0
  Death | 0

4. Primary Outcome: Number of Participants With Clinically Significant Abnormalities in Vital Signs
Description: Vital signs parameters included blood pressure (hypotension and hypertension), pulse rate (tachycardia and bradycardia), body temperature and respiratory rate. Any change in vital sign abnormalities that was clinically significant in the medical and scientific judgment of the investigator and not related to an underlying disease was reported as an unsolicited adverse event (AE). Any clinically significant abnormality associated with underlying disease does not require reporting as an (S)AE unless judged by the investigator to be more severe than expected for the participant's condition.
Time Frame: During first hour post vaccination (vaccine administered at Day 1)
Population: The analysis was performed on the Safety Analysis Set which consisted of all randomized participants who received a vaccination in this study with either ASP3772, PCV13, or PPSV23.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1, Group 1 Adults, ASP3772 Low Dose | Stage 1, Group 1 Adults, ASP3772 Medium Dose | Stage 1, Group 1 Adults, ASP3772 High Dose | Stage 1, Group 1, PCV13 Pooled Comparator | Stage 2, Group 2 Older Adults, ASP3772 Low Dose | Stage 2, Group 2 Older Adults, ASP3772 Medium Dose | Stage 2, Group 2 Older Adults, ASP3772 High Dose | Stage 2, Group 2, PCV13 Pooled Comparator | Stage 2, Group 3, PPSV23 Comparator
Number analyzed (Participants) | 30 | 31 | 32 | 33 | 100 | 107 | 86 | 97 | 113
Participants
  Temperature Increase | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Tachycardia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Bradycardia | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Hypertension (systolic) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0
  Hypertension (diastolic) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Hypotension (systolic) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Respiratory Rate | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 3 | 0

5. Primary Outcome: Number of Participants With Potentially Clinically Significant Laboratory Values
Description: Clinical laboratory testing included hematology, clinical chemistry, or urinalysis. Any abnormal laboratory test result (e.g., in hematology, clinical chemistry, or urinalysis) that was clinically significant in the medical and scientific judgment of the investigator and not related to an underlying disease was reported as an unsolicited adverse event (AE). Laboratory tests of clinical interest included total bilirubin ≥ 2x ULN and Alkaline phosphatase > 1.5 × upper limit of normal. Study Investigator's interest was to assess only potentially clinically significant values.
Time Frame: Up to Day 30
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Groups:
- Stage 2, Group 3, PPSV23 Comparato: Older adults aged 65 to 85 years, who had previously been previously vaccinated with PCV13, were enrolled and received a single of dose PPSV23 on Day 1.
  113
Arm/Group | Stage 1, Group 1 Adults, ASP3772 Low Dose | Stage 1, Group 1 Adults, ASP3772 Medium Dose | Stage 1, Group 1 Adults, ASP3772 High Dose | Stage 1, Group 1, PCV13 Pooled Comparator | Stage 2, Group 2 Older Adults, ASP3772 Low Dose | Stage 2, Group 2 Older Adults, ASP3772 Medium Dose | Stage 2, Group 2 Older Adults, ASP3772 High Dose | Stage 2, Group 2, PCV13 Pooled Comparator | Stage 2, Group 3, PPSV23 Comparato
Number analyzed (Participants) | 30 | 31 | 32 | 33 | 100 | 107 | 86 | 97 | 113
Participants
  Total Bilirubin: number analyzed (Participants) | 30 | 31 | 32 | 33 | 100 | 107 | 86 | 95 | 113
  Total Bilirubin | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Alkaline phosphatase: number analyzed (Participants) | 30 | 31 | 32 | 33 | 100 | 107 | 86 | 96 | 113
  Alkaline phosphatase | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

6. Primary Outcome: Number of Participants With Potentially Clinically Significant Physical Examination Values
Description: A physical examination consists of an examination of general appearance, eyes, nose throat, neck (including thyroid), lymph nodes, chest, lungs, cardiovascular, abdomen, skin, extremities, musculoskeletal and neurological system including mental status. Any abnormal test result that was clinically significant in the medical and scientific judgment of the investigator and not related to an underlying disease was reported as an unsolicited adverse event (AE). Study Investigator's interest was to assess only potentially clinically significant values.
Time Frame: Up to Day 30
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1, Group 1 Adults, ASP3772 Low Dose | Stage 1, Group 1 Adults, ASP3772 Medium Dose | Stage 1, Group 1 Adults, ASP3772 High Dose | Stage 1, Group 1, PCV13 Pooled Comparator | Stage 2, Group 2 Older Adults, ASP3772 Low Dose | Stage 2, Group 2 Older Adults, ASP3772 Medium Dose | Stage 2, Group 2 Older Adults, ASP3772 High Dose | Stage 2, Group 2, PCV13 Pooled Comparator | Stage 2, Group 3, PPSV23 Comparato
Number analyzed (Participants) | 30 | 31 | 32 | 33 | 100 | 107 | 86 | 97 | 113
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Number of Participants With Clinically Significant Abnormal Electrocardiogram (ECG), [Stage 1, Group 1] and [Stage 2, Group 2]
Description: The Investigator assessed standard 12-lead ECG recordings for the purposes of safety assessment and participant management.
  Any clinically significant abnormality, as determined by the investigator's medical and scientific judgment and unrelated to underlying disease, should be reported as an unsolicited (S)AE.
  Any clinically significant abnormality associated with underlying disease does not require reporting as an (S)AE unless judged by the investigator to be more severe than expected for the participant's condition.
Time Frame: Day - 28 to Day -1 (28 days prior to study vaccination)
Population: The analysis was performed on the Safety Analysis Set which consisted of all randomized participants who received a vaccination in this study with either ASP3772 or PCV13 and for whom ECG data was available at Day -28 to Day -1.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1, Group 1 Adults, ASP3772 Low Dose | Stage 1, Group 1 Adults, ASP3772 Medium Dose | Stage 1, Group 1 Adults, ASP3772 High Dose | Stage 1, Group 1, PCV13 Pooled Comparator | Stage 2, Group 2 Older Adults, ASP3772 Low Dose | Stage 2, Group 2 Older Adults, ASP3772 Medium Dose | Stage 2, Group 2 Older Adults, ASP3772 High Dose | Stage 2, Group 2, PCV13 Pooled Comparator
Number analyzed (Participants) | 30 | 31 | 32 | 33 | 98 | 107 | 76 | 92
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: Number of Participants With Clinically Significant Abnormal Electrocardiogram (ECG), [Stage 1, Group 1] and [Stage 2, Group 2]
Description: as for outcome 7
Time Frame: At Day 7
Population: The analysis was performed on the Safety Analysis Set which consisted of all randomized participants who received a vaccination in this study with either ASP3772 or PCV13 and for whom ECG data was available at Day 7.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1, Group 1 Adults, ASP3772 Low Dose | Stage 1, Group 1 Adults, ASP3772 Medium Dose | Stage 1, Group 1 Adults, ASP3772 High Dose | Stage 1, Group 1, PCV13 Pooled Comparator | Stage 2, Group 2 Older Adults, ASP3772 Low Dose | Stage 2, Group 2 Older Adults, ASP3772 Medium Dose | Stage 2, Group 2 Older Adults, ASP3772 High Dose | Stage 2, Group 2, PCV13 Pooled Comparator
Number analyzed (Participants) | 30 | 30 | 32 | 33 | 95 | 106 | 86 | 93
Participants | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0

9. Primary Outcome: Number of Participants With Clinically Significant Abnormal Electrocardiogram (ECG), [Stage 2, Group 3]
Description: as for outcome 7
Time Frame: Day - 28 to Day -1 (28 days prior to study vaccination)
Population: The analysis was performed on the Safety Analysis Set which consisted of all enrolled participants in Stage 2, Group 3 who received a vaccination in this study with PPSV23 and for whom ECG data was available at Day -28 to Day -1.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2, Group 3, PPSV23 Comparator
Number analyzed (Participants) | 108
Participants | 0

10. Primary Outcome: Reactogenicity Assessed by Number of Participants With Solicited Local Reactions, [Stage 1, Group 1]
Description: Local reactions include pain, tenderness, redness/erythema, swelling and induration.
Time Frame: Up to 7 Day post Vaccination (vaccine administered at Day 1)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1, Group 1 Adults, ASP3772 Low Dose | Stage 1, Group 1 Adults, ASP3772 Medium Dose | Stage 1, Group 1 Adults, ASP3772 High Dose | Stage 1, Group 1, PCV13 Pooled Comparator
Number analyzed (Participants) | 30 | 31 | 32 | 33
Participants
  Tenderness | 15 | 22 | 20 | 25
  Pain | 16 | 19 | 20 | 24
  Induration | 0 | 2 | 1 | 4
  Erythema/Redness | 0 | 2 | 0 | 3
  Swelling | 0 | 1 | 0 | 3

11. Primary Outcome: Reactogenicity Assessed by Number of Solicited Local Reactions, [Stage 2, Group 2 and Group 3]
Description: Assessed solicited local reactions were pain, tenderness, redness/erythema, swelling, induration, itching at injection site and pruritus at injection site.
Time Frame: Up to 7 Day post Vaccination (vaccine administered at Day 1)
Population: The analysis was performed on the Safety Analysis Set which consisted of all randomized participants who received a vaccination in this study with either ASP3772 or PPSV23.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2, Group 2 Older Adults, ASP3772 Low Dose | Stage 2, Group 2 Older Adults, ASP3772 Medium Dose | Stage 2, Group 2 Older Adults, ASP3772 High Dose | Stage 2, Group 2, PCV13 Pooled Comparator | Stage 2, Group 3, PPSV23 Comparator
Number analyzed (Participants) | 100 | 107 | 86 | 97 | 113
Participants
  Tenderness | 38 | 51 | 48 | 42 | 0
  Pain | 26 | 37 | 38 | 33 | 0
  Induration | 2 | 6 | 4 | 2 | 0
  Erythema/Redness | 1 | 4 | 5 | 4 | 0
  Swelling | 1 | 6 | 3 | 4 | 0
  Other Illness/Clinical Event-Itching At Injection Site | 0 | 1 | 0 | 0 | 0
  Other Illness/Clinical Event-Pruritus At Injection Site | 0 | 0 | 0 | 1 | 0

12. Primary Outcome: Reactogenicity Assessed by Number of Solicited Systemic Reactions, [Stage 1, Group 1]
Description: Assessed systemic reactions were nausea/vomiting, diarrhea, headache, fever, fatigue and muscle discomfort or pain/myalgia.
Time Frame: Up to 7 Day post Vaccination (vaccine administered at Day 1)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1, Group 1 Adults, ASP3772 Low Dose | Stage 1, Group 1 Adults, ASP3772 Medium Dose | Stage 1, Group 1 Adults, ASP3772 High Dose | Stage 1, Group 1, PCV13 Pooled Comparator
Number analyzed (Participants) | 30 | 31 | 32 | 33
Participants
  Fatigue | 7 | 8 | 10 | 13
  Myalgia | 7 | 7 | 11 | 13
  Headache | 5 | 6 | 7 | 13
  Diarrhea | 4 | 2 | 4 | 6
  Nausea | 3 | 5 | 2 | 3
  Fever | 0 | 3 | 1 | 0
  Vomiting | 0 | 1 | 1 | 1

13. Primary Outcome: Reactogenicity Assessed by Number of Solicited Systemic Reactions [Stage 2, Group 2 and Group 3]
Description: as for outcome 12
Time Frame: Up to 7 Day post Vaccination (vaccine administered at Day 1)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2, Group 2 Older Adults, ASP3772 Low Dose | Stage 2, Group 2 Older Adults, ASP3772 Medium Dose | Stage 2, Group 2 Older Adults, ASP3772 High Dose | Stage 2, Group 2, PCV13 Pooled Comparator | Stage 2, Group 3, PPSV23 Comparator
Number analyzed (Participants) | 100 | 107 | 86 | 97 | 113
Participants
  Myalgia | 11 | 26 | 27 | 17 | 0
  Fatigue | 18 | 18 | 22 | 21 | 0
  Headache | 13 | 12 | 10 | 10 | 0
  Diarrhea | 3 | 15 | 13 | 6 | 0
  Arthralgia | 5 | 10 | 13 | 8 | 0
  Nausea | 4 | 9 | 2 | 6 | 0
  Vomiting | 1 | 1 | 1 | 2 | 0

14. Secondary Outcome: Geometric Mean Titers (GMTs) for Serotype-specific Opsonophagocytic Activity (OPA) Titer, [Stage 1, Group 1]
Description: OPA titers were determined for serotypes: 1, 3,4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F. OPA titer was expressed as the reciprocal of the serum dilution that causes a 50% reduction in the colony-forming units.
Time Frame: At Day 1 and Day 30
Population: The analysis was performed on the Full Analysis Set which consisted of all randomized Participants who received a vaccination in this study with either ASP3772 or PCV13, had at least 1 post vaccination measurement and for whom immunogenicity data was collected for specific serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Stage 1, Group 1 Adults, ASP3772 Low Dose | Stage 1, Group 1 Adults, ASP3772 Medium Dose | Stage 1, Group 1 Adults, ASP3772 High Dose | Stage 1, Group 1, PCV13 Pooled Comparator
Number analyzed (Participants) | 29 | 31 | 32 | 33
Titers
  Serotype 1, Day 1: number analyzed (Participants) | 29 | 30 | 32 | 32
  Serotype 1, Day 1 | 7.5 [5.2 to 10.7] | 7.6 [5.3 to 10.9] | 7.7 [5.6 to 10.6] | 6.5 [4.6 to 9.2]
  Serotype 1, Day 30: number analyzed (Participants) | 29 | 29 | 31 | 31
  Serotype 1, Day 30 | 448.4 [298.4 to 673.7] | 347.0 [239.0 to 503.7] | 337.6 [204.4 to 557.7] | 482.1 [295.1 to 787.5]
  Serotype 3, Day 1: number analyzed (Participants) | 27 | 19 | 25 | 29
  Serotype 3, Day 1 | 33.5 [17.7 to 63.4] | 43.6 [22.2 to 85.5] | 14.4 [8.3 to 24.9] | 21.4 [12.0 to 37.9]
  Serotype 3, Day 30: number analyzed (Participants) | 28 | 26 | 16 | 24
  Serotype 3, Day 30 | 368.1 [276.2 to 490.6] | 485.7 [394.1 to 598.6] | 432.6 [306.4 to 610.7] | 337.7 [221.1 to 515.8]
  Serotype 4, Day 1: number analyzed (Participants) | 26 | 25 | 22 | 25
  Serotype 4, Day 1 | 46.8 [15.9 to 137.2] | 29.4 [11.5 to 75.7] | 77.1 [29.7 to 200.2] | 42.2 [16.0 to 111.5]
  Serotype 4, Day 30: number analyzed (Participants) | 29 | 27 | 25 | 29
  Serotype 4, Day 30 | 4038.7 [3141.8 to 5191.8] | 2452.8 [1359.9 to 4424.1] | 5211.8 [3483.0 to 7798.7] | 4912.1 [3183.9 to 7578.3]
  Serotype 5, Day 1: number analyzed (Participants) | 29 | 31 | 32 | 32
  Serotype 5, Day 1 | 12.5 [5.7 to 27.5] | 8.0 [4.9 to 13] | 6.1 [4.4 to 8.5] | 6.6 [4.0 to 10.7]
  Serotype 5, Day 30: number analyzed (Participants) | 29 | 29 | 31 | 31
  Serotype 5, Day 30 | 1344.0 [930.1 to 1942.0] | 1193.9 [675.3 to 2110.9] | 1557.3 [1092.0 to 2220.9] | 1954.8 [1337.9 to 2856.0]
  Serotype 6A, Day1: number analyzed (Participants) | 27 | 29 | 29 | 30
  Serotype 6A, Day1 | 64.3 [26.4 to 156.7] | 55.8 [26.4 to 118.2] | 78.6 [32.7 to 188.7] | 76.5 [32.5 to 180.2]
  Serotype 6A, Day 30: number analyzed (Participants) | 28 | 29 | 31 | 30
  Serotype 6A, Day 30 | 9817.6 [6133.9 to 15713.3] | 6018.5 [3213.3 to 11272.6] | 6953.5 [4675.5 to 10341.6] | 18733.9 [12189.2 to 28792.5]
  Serotype 6B, Day 1: number analyzed (Participants) | 28 | 29 | 29 | 28
  Serotype 6B, Day 1 | 110.1 [39.8 to 304.9] | 119.8 [56.3 to 255.0] | 65.7 [32.7 to 131.7] | 92.3 [38.1 to 223.4]
  Serotype 6B, Day 30: number analyzed (Participants) | 29 | 26 | 28 | 27
  Serotype 6B, Day 30 | 7742.8 [5776.7 to 10378.0] | 4981.0 [3211.1 to 7726.5] | 4720.9 [3214.1 to 6934.0] | 10986.7 [7116.4 to 16962.0]
  Serotype 7F, Day 1: number analyzed (Participants) | 24 | 30 | 28 | 28
  Serotype 7F, Day 1 | 1003.2 [392.4 to 2565.0] | 422.8 [171.1 to 1044.9] | 412.5 [154.5 to 1101.2] | 1325.5 [790.4 to 2222.7]
  Serotype 7F, Day 30: number analyzed (Participants) | 29 | 29 | 30 | 29
  Serotype 7F, Day 30 | 7185.5 [5104.6 to 10114.7] | 6025.6 [4913.8 to 7388.9] | 7223.4 [5417.6 to 9631.0] | 8855.7 [6388.9 to 12274.9]
  Serotype 9V, Day 1: number analyzed (Participants) | 29 | 31 | 31 | 31
  Serotype 9V, Day 1 | 1106.5 [605.1 to 2023.5] | 279.4 [107.4 to 727.2] | 360.9 [156.0 to 834.8] | 577.6 [268.2 to 1243.8]
  Serotype 9V, Day 30: number analyzed (Participants) | 29 | 29 | 31 | 30
  Serotype 9V, Day 30 | 8458.4 [5783.2 to 12371.0] | 7789.6 [5051.3 to 12012.4] | 10532.3 [7817.6 to 14189.7] | 13756.2 [8965.1 to 21107.5]
  Serotype 14, Day 1: number analyzed (Participants) | 26 | 27 | 27 | 30
  Serotype 14, Day 1 | 592.9 [257.1 to 1367.2] | 269.7 [111.8 to 650.8] | 138.2 [45.4 to 421.0] | 141.1 [51.6 to 385.7]
  Serotype 14, Day 30: number analyzed (Participants) | 29 | 29 | 31 | 31
  Serotype 14, Day 30 | 5407.3 [3328.8 to 8783.7] | 2805.5 [1161.4 to 6776.9] | 11292.9 [6725.4 to 18962.5] | 9982.6 [6004.5 to 16596.4]
  Serotype 18C, Day 1: number analyzed (Participants) | 29 | 30 | 30 | 30
  Serotype 18C, Day 1 | 74.7 [28.8 to 193.8] | 119.3 [53.4 to 266.5] | 123.0 [54.0 to 280.5] | 100.6 [42.3 to 239.2]
  Serotype 18C, Day 30: number analyzed (Participants) | 29 | 28 | 31 | 31
  Serotype 18C, Day 30 | 6779.7 [4488.1 to 10241.5] | 5266.3 [3253.8 to 8523.6] | 6077.0 [4315.7 to 8557.2] | 7592.1 [5455.2 to 10565.9]
  Serotype 19A, Day 1: number analyzed (Participants) | 28 | 29 | 30 | 32
  Serotype 19A, Day 1 | 732.8 [411.7 to 1304.1] | 469.0 [250.3 to 878.9] | 489.9 [306.7 to 782.6] | 657.8 [374.3 to 1156.1]
  Serotype 19A, Day 30: number analyzed (Participants) | 28 | 28 | 31 | 30
  Serotype 19A, Day 30 | 3879.0 [2750.8 to 5469.8] | 5357.2 [3802.0 to 7548.5] | 4866.3 [3601.4 to 6575.5] | 7695.1 [5705.5 to 10378.5]
  Serotype 19F, Day 1: number analyzed (Participants) | 29 | 29 | 31 | 31
  Serotype 19F, Day 1 | 221.4 [93.2 to 525.9] | 391.4 [176.2 to 869.3] | 457.9 [247.7 to 846.5] | 316.0 [157.1 to 635.6]
  Serotype 19F, Day 30: number analyzed (Participants) | 29 | 29 | 31 | 31
  Serotype 19F, Day 30 | 3397.2 [2572.4 to 4486.4] | 3862.5 [2682.0 to 5562.7] | 5636.2 [4136.8 to 7679.0] | 6065.2 [3976.2 to 9251.5]
  Serotype 23F, Day 1: number analyzed (Participants) | 23 | 21 | 21 | 20
  Serotype 23F, Day 1 | 230.6 [71.3 to 745.7] | 141.0 [49.4 to 402.4] | 69.9 [24.0 to 203.9] | 103.9 [33.9 to 318.5]
  Serotype 23F, Day 30: number analyzed (Participants) | 28 | 22 | 21 | 27
  Serotype 23F, Day 30 | 2947.8 [1490.1 to 5831.7] | 2951.1 [1464.8 to 5945.5] | 3399.7 [1569.3 to 7364.7] | 15054.3 [8573.2 to 26435.0]
Statistical Analysis 1: Comparison: Stage 1, Group 1 Adults, ASP3772 Low Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 1, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.14, 95% CI 2-sided [0.70 to 1.85]
Statistical Analysis 2: Comparison: Stage 1, Group 1 Adults, ASP3772 Medium Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 1, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.17, 95% CI 2-sided [0.72 to 1.90]
Statistical Analysis 3: Comparison: Stage 1, Group 1 Adults, ASP3772 High Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 1, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.17, 95% CI 2-sided [0.74 to 1.87]
Statistical Analysis 4: Comparison: Stage 1, Group 1 Adults, ASP3772 Low Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 3, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.57, 95% CI 2-sided [0.68 to 3.63]
Statistical Analysis 5: Comparison: Stage 1, Group 1 Adults, ASP3772 Medium Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 3, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 2.04, 95% CI 2-sided [0.86 to 4.82]
Statistical Analysis 6: Comparison: Stage 1, Group 1 Adults, ASP3772 High Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 3, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.67, 95% CI 2-sided [0.31 to 1.46]
Statistical Analysis 7: Comparison: Stage 1, Group 1 Adults, ASP3772 Low Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 4, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.11, 95% CI 2-sided [0.27 to 4.55]
Statistical Analysis 8: Comparison: Stage 1, Group 1 Adults, ASP3772 Medium Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 4, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.70, 95% CI 2-sided [0.19 to 2.61]
Statistical Analysis 9: Comparison: Stage 1, Group 1 Adults, ASP3772 High Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 4, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.83, 95% CI 2-sided [0.49 to 6.85]
Statistical Analysis 10: Comparison: Stage 1, Group 1 Adults, ASP3772 Low Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 5, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.90, 95% CI 2-sided [0.76 to 4.73]
Statistical Analysis 11: Comparison: Stage 1, Group 1 Adults, ASP3772 Medium Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 5, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.22, 95% CI 2-sided [0.62 to 2.40]
Statistical Analysis 12: Comparison: Stage 1, Group 1 Adults, ASP3772 High Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 5, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.93, 95% CI 2-sided [0.52 to 1.65]
Statistical Analysis 13: Comparison: Stage 1, Group 1 Adults, ASP3772 Low Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 6A, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.84, 95% CI 2-sided [0.25 to 2.82]
Statistical Analysis 14: Comparison: Stage 1, Group 1 Adults, ASP3772 Medium Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 6A, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.73, 95% CI 2-sided [0.24 to 2.23]
Statistical Analysis 15: Comparison: Stage 1, Group 1 Adults, ASP3772 High Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 6A, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.03, 95% CI 2-sided [0.31 to 3.41]
Statistical Analysis 16: Comparison: Stage 1, Group 1 Adults, ASP3772 Low Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 6B,Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.19, 95% CI 2-sided [0.32 to 4.46]
Statistical Analysis 17: Comparison: Stage 1, Group 1 Adults, ASP3772 Medium Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 6B, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.30, 95% CI 2-sided [0.42 to 4.05]
Statistical Analysis 18: Comparison: Stage 1, Group 1 Adults, ASP3772 High Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 6B, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.71, 95% CI 2-sided [0.24 to 2.14]
Statistical Analysis 19: Comparison: Stage 1, Group 1 Adults, ASP3772 Low Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 7F, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.76, 95% CI 2-sided [0.26 to 2.17]
Statistical Analysis 20: Comparison: Stage 1, Group 1 Adults, ASP3772 Medium Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 7F, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.32, 95% CI 2-sided [0.11 to 0.89]
Statistical Analysis 21: Comparison: Stage 1, Group 1 Adults, ASP3772 High Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 7F, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.31, 95% CI 2-sided [0.10 to 0.93]
Statistical Analysis 22: Comparison: Stage 1, Group 1 Adults, ASP3772 Low Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 9V, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.92, 95% CI 2-sided [0.74 to 4.99]
Statistical Analysis 23: Comparison: Stage 1, Group 1 Adults, ASP3772 Medium Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 9V, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.48, 95% CI 2-sided [0.15 to 1.61]
Statistical Analysis 24: Comparison: Stage 1, Group 1 Adults, ASP3772 High Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 9V, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.62, 95% CI 2-sided [0.21 to 1.90]
Statistical Analysis 25: Comparison: Stage 1, Group 1 Adults, ASP3772 Low Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 14, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 4.20, 95% CI 2-sided [1.17 to 15.09]
Statistical Analysis 26: Comparison: Stage 1, Group 1 Adults, ASP3772 Medium Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 14, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.91, 95% CI 2-sided [0.52 to 7.07]
Statistical Analysis 27: Comparison: Stage 1, Group 1 Adults, ASP3772 High Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 14, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.98, 95% CI 2-sided [0.23 to 4.25]
Statistical Analysis 28: Comparison: Stage 1, Group 1 Adults, ASP3772 Low Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 18C, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.74, 95% CI 2-sided [0.21 to 2.62]
Statistical Analysis 29: Comparison: Stage 1, Group 1 Adults, ASP3772 Medium Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 18C, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.19, 95% CI 2-sided [0.37 to 3.77]
Statistical Analysis 30: Comparison: Stage 1, Group 1 Adults, ASP3772 High Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 18C, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.22, 95% CI 2-sided [0.38 to 3.94]
Statistical Analysis 31: Comparison: Stage 1, Group 1 Adults, ASP3772 Low Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 19A, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.11, 95% CI 2-sided [0.51 to 2.45]
Statistical Analysis 32: Comparison: Stage 1, Group 1 Adults, ASP3772 Medium Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 19A, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.71, 95% CI 2-sided [0.31 to 1.63]
Statistical Analysis 33: Comparison: Stage 1, Group 1 Adults, ASP3772 High Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 19A, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.74, 95% CI 2-sided [0.36 to 1.53]
Statistical Analysis 34: Comparison: Stage 1, Group 1 Adults, ASP3772 Low Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 19F, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.70, 95% CI 2-sided [0.24 to 2.08]
Statistical Analysis 35: Comparison: Stage 1, Group 1 Adults, ASP3772 Medium Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 19F, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.24, 95% CI 2-sided [0.44 to 3.50]
Statistical Analysis 36: Comparison: Stage 1, Group 1 Adults, ASP3772 High Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 19F, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.45, 95% CI 2-sided [0.58 to 3.61]
Statistical Analysis 37: Comparison: Stage 1, Group 1 Adults, ASP3772 Low Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 23F, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 2.22, 95% CI 2-sided [0.46 to 10.69]
Statistical Analysis 38: Comparison: Stage 1, Group 1 Adults, ASP3772 Medium Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 23F, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.36, 95% CI 2-sided [0.31 to 5.99]
Statistical Analysis 39: Comparison: Stage 1, Group 1 Adults, ASP3772 High Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 23F, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.67, 95% CI 2-sided [0.15 to 3.01]
Statistical Analysis 40: Comparison: Stage 1, Group 1 Adults, ASP3772 Low Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 1, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.93, 95% CI 2-sided [0.50 to 1.74]
Statistical Analysis 41: Comparison: Stage 1, Group 1 Adults, ASP3772 Medium Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 1, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.72, 95% CI 2-sided [0.39 to 1.32]
Statistical Analysis 42: Comparison: Stage 1, Group 1 Adults, ASP3772 High Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 1, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.70, 95% CI 2-sided [0.35 to 1.39]
Statistical Analysis 43: Comparison: Stage 1, Group 1 Adults, ASP3772 Low Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 3, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.09, 95% CI 2-sided [0.66 to 1.80]
Statistical Analysis 44: Comparison: Stage 1, Group 1 Adults, ASP3772 Medium Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 3, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.44, 95% CI 2-sided [0.90 to 2.29]
Statistical Analysis 45: Comparison: Stage 1, Group 1 Adults, ASP3772 High Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 3, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.28, 95% CI 2-sided [0.76 to 2.17]
Statistical Analysis 46: Comparison: Stage 1, Group 1 Adults, ASP3772 Low Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 4, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.82, 95% CI 2-sided [0.50 to 1.35]
Statistical Analysis 47: Comparison: Stage 1, Group 1 Adults, ASP3772 Medium Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 4, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.50, 95% CI 2-sided [0.24 to 1.02]
Statistical Analysis 48: Comparison: Stage 1, Group 1 Adults, ASP3772 High Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 4, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.06, 95% CI 2-sided [0.60 to 1.89]
Statistical Analysis 49: Comparison: Stage 1, Group 1 Adults, ASP3772 Low Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 5, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.69, 95% CI 2-sided [0.41 to 1.15]
Statistical Analysis 50: Comparison: Stage 1, Group 1 Adults, ASP3772 Medium Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 5, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.61, 95% CI 2-sided [0.31 to 1.20]
Statistical Analysis 51: Comparison: Stage 1, Group 1 Adults, ASP3772 High Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 5, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.80, 95% CI 2-sided [0.48 to 1.32]
Statistical Analysis 52: Comparison: Stage 1, Group 1 Adults, ASP3772 Low Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 6A, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.52, 95% CI 2-sided [0.28 to 0.98]
Statistical Analysis 53: Comparison: Stage 1, Group 1 Adults, ASP3772 Medium Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 6A, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.32, 95% CI 2-sided [0.15 to 0.68]
Statistical Analysis 54: Comparison: Stage 1, Group 1 Adults, ASP3772 High Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 6A, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.37, 95% CI 2-sided [0.21 to 0.66]
Statistical Analysis 55: Comparison: Stage 1, Group 1 Adults, ASP3772 Low Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 6B, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.70, 95% CI 2-sided [0.42 to 1.18]
Statistical Analysis 56: Comparison: Stage 1, Group 1 Adults, ASP3772 Medium Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 6B, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.45, 95% CI 2-sided [0.25 to 0.83]
Statistical Analysis 57: Comparison: Stage 1, Group 1 Adults, ASP3772 High Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 6B, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.43, 95% CI 2-sided [0.24 to 0.76]
Statistical Analysis 58: Comparison: Stage 1, Group 1 Adults, ASP3772 Low Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 7F, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.81, 95% CI 2-sided [0.51 to 1.29]
Statistical Analysis 59: Comparison: Stage 1, Group 1 Adults, ASP3772 Medium Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 7F, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.68, 95% CI 2-sided [0.47 to 0.99]
Statistical Analysis 60: Comparison: Stage 1, Group 1 Adults, ASP3772 High Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 7F, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.82, 95% CI 2-sided [0.53 to 1.25]
Statistical Analysis 61: Comparison: Stage 1, Group 1 Adults, ASP3772 Low Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 9V, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.61, 95% CI 2-sided [0.35 to 1.08]
Statistical Analysis 62: Comparison: Stage 1, Group 1 Adults, ASP3772 Medium Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 9V, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.57, 95% CI 2-sided [0.31 to 1.03]
Statistical Analysis 63: Comparison: Stage 1, Group 1 Adults, ASP3772 High Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 9V, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.77, 95% CI 2-sided [0.46 to 1.28]
Statistical Analysis 64: Comparison: Stage 1, Group 1 Adults, ASP3772 Low Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 14, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.54, 95% CI 2-sided [0.27 to 1.08]
Statistical Analysis 65: Comparison: Stage 1, Group 1 Adults, ASP3772 Medium Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 14, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.28, 95% CI 2-sided [0.10 to 0.77]
Statistical Analysis 66: Comparison: Stage 1, Group 1 Adults, ASP3772 High Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 14, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.13, 95% CI 2-sided [0.56 to 2.30]
Statistical Analysis 67: Comparison: Stage 1, Group 1 Adults, ASP3772 Low Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 18C, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.89, 95% CI 2-sided [0.53 to 1.50]
Statistical Analysis 68: Comparison: Stage 1, Group 1 Adults, ASP3772 Medium Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 18C, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.69, 95% CI 2-sided [0.39 to 1.23]
Statistical Analysis 69: Comparison: Stage 1, Group 1 Adults, ASP3772 High Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 18C, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.80, 95% CI 2-sided [0.50 to 1.28]
Statistical Analysis 70: Comparison: Stage 1, Group 1 Adults, ASP3772 Low Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 19A, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.50, 95% CI 2-sided [0.32 to 0.79]
Statistical Analysis 71: Comparison: Stage 1, Group 1 Adults, ASP3772 Medium Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 19A, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.70, 95% CI 2-sided [0.45 to 1.09]
Statistical Analysis 72: Comparison: Stage 1, Group 1 Adults, ASP3772 High Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 19A, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.63, 95% CI 2-sided [0.42 to 0.96]
Statistical Analysis 73: Comparison: Stage 1, Group 1 Adults, ASP3772 Low Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 19F, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.56, 95% CI 2-sided [0.34 to 0.92]
Statistical Analysis 74: Comparison: Stage 1, Group 1 Adults, ASP3772 Medium Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 19F, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.64, 95% CI 2-sided [0.37 to 1.10]
Statistical Analysis 75: Comparison: Stage 1, Group 1 Adults, ASP3772 High Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 19F, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.93, 95% CI 2-sided [0.56 to 1.55]
Statistical Analysis 76: Comparison: Stage 1, Group 1 Adults, ASP3772 Low Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 23F, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.20, 95% CI 2-sided [0.08 to 0.46]
Statistical Analysis 77: Comparison: Stage 1, Group 1 Adults, ASP3772 Medium Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 23F, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.20, 95% CI 2-sided [0.08 to 0.47]
Statistical Analysis 78: Comparison: Stage 1, Group 1 Adults, ASP3772 High Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 23F, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.23, 95% CI 2-sided [0.09 to 0.57]

15. Secondary Outcome: Geometric Mean Concentration (GMCs) for Serotype-specific Immunoglobulin G (IgG), [Stage 1, Group 1]
Description: Immunological responses were assessed in terms of IgG GMCs and expressed as titers. The assessed serotypes were: 1, 3,4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F.
Time Frame: At Day 1 and Day 30
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Stage 1, Group 1 Adults, ASP3772 Low Dose | Stage 1, Group 1 Adults, ASP3772 Medium Dose | Stage 1, Group 1 Adults, ASP3772 High Dose | Stage 1, Group 1, PCV13 Pooled Comparator
Number analyzed (Participants) | 30 | 31 | 32 | 33
Titers
  Serotype 1, Day 1 | 190.4 [110.0 to 329.8] | 177.2 [109.8 to 285.9] | 252.8 [156.1 to 409.3] | 177.1 [107.0 to 293.1]
  Serotype 1, Day 30: number analyzed (Participants) | 29 | 30 | 31 | 32
  Serotype 1, Day 30 | 5174.8 [3459.5 to 7740.6] | 7023.9 [4786.0 to 10308.2] | 11097.1 [7934.9 to 15519.5] | 7407.4 [4595.0 to 11941.2]
  Serotype 3, Day 1 | 103.7 [57.3 to 187.6] | 135.9 [92.4 to 199.9] | 101.6 [70.6 to 146.3] | 82.2 [50.3 to 134.1]
  Serotype 3, Day 30: number analyzed (Participants) | 30 | 30 | 31 | 32
  Serotype 3, Day 30 | 755.8 [519.3 to 1100.0] | 1465.6 [1088.8 to 1972.8] | 2115.7 [1571.6 to 2848.1] | 547.0 [386.4 to 774.2]
  Serotype 4, Day 1 | 85.6 [50.5 to 144.8] | 68.5 [39.8 to 117.9] | 103.2 [61.4 to 173.6] | 83.4 [48.4 to 143.7]
  Serotype 4, Day 30: number analyzed (Participants) | 30 | 30 | 31 | 32
  Serotype 4, Day 30 | 2709.5 [1827.5 to 4017.3] | 2171.4 [1508.5 to 3125.6] | 4778.6 [3114.7 to 7331.4] | 2129.3 [1348.0 to 3363.4]
  Serotype 5, Day 1 | 194.6 [101.5 to 373.2] | 82.0 [50.8 to 132.2] | 105.5 [67.4 to 165.0] | 113.8 [66.6 to 194.7]
  Serotype 5, Day 30: number analyzed (Participants) | 30 | 30 | 31 | 32
  Serotype 5, Day 30 | 7426.7 [4829.4 to 11420.8] | 3946.3 [2228.0 to 6989.8] | 6973.3 [4416.2 to 11011.0] | 4691.0 [2318.4 to 9491.4]
  Serotype 6A, Day 1 | 192.8 [115.3 to 322.5] | 206.8 [134.6 to 317.7] | 175.9 [106.8 to 289.6] | 161.5 [92.0 to 283.6]
  Serotype 6A, Day 30: number analyzed (Participants) | 30 | 30 | 31 | 32
  Serotype 6A, Day 30 | 8735.6 [5103.5 to 14952.5] | 7585.4 [4028.4 to 14283.4] | 6805.0 [4084.3 to 11338.0] | 9819.2 [5487.6 to 17569.8]
  Serotype 6B, Day 1 | 199.6 [99.5 to 400.4] | 155.9 [93.0 to 261.3] | 130.7 [82.7 to 206.6] | 162.4 [86.2 to 305.9]
  Serotype 6B, Day 30: number analyzed (Participants) | 30 | 30 | 31 | 32
  Serotype 6B, Day 30 | 14638.6 [8712.2 to 24596.4] | 8728.4 [4656.8 to 16360.1] | 10206.8 [6083.2 to 17125.7] | 11576.4 [6130.6 to 21860.0]
  Serotype 7F, Day 1 | 305.8 [170.1 to 549.7] | 234.5 [164.0 to 335.4] | 342.6 [230.0 to 510.2] | 202.8 [137.9 to 298.3]
  Serotype 7F, Day 30: number analyzed (Participants) | 30 | 30 | 31 | 32
  Serotype 7F, Day 30 | 7131.3 [4960.4 to 10252.4] | 7580.7 [5169.8 to 11115.9] | 11037.5 [7653.3 to 15918.1] | 3830.9 [2423.0 to 6056.8]
  Serotype 9V, Day 1 | 152.7 [90.7 to 257.0] | 104.2 [73.2 to 148.3] | 119.4 [85.1 to 167.6] | 139.9 [84.8 to 230.7]
  Serotype 9V, Day 30: number analyzed (Participants) | 30 | 30 | 31 | 32
  Serotype 9V, Day 30 | 3791.8 [2479.8 to 5797.8] | 5523.5 [3890.7 to 7841.4] | 6681.5 [4440.9 to 10052.6] | 3968.6 [2312.1 to 6811.7]
  Serotype 14, Day 1 | 837.6 [423.6 to 1656.1] | 1062.2 [582.1 to 1938.4] | 363.8 [186.7 to 708.9] | 408.7 [224.0 to 745.7]
  Serotype 14, Day 30: number analyzed (Participants) | 30 | 30 | 31 | 32
  Serotype 14, Day 30 | 16115.3 [8502.1 to 30545.5] | 17185.4 [9582.7 to 30820.1] | 33150.4 [18372.0 to 59816.3] | 15893.1 [8049.8 to 31378.2]
  Serotype 18C, Day 1 | 282.4 [151.5 to 526.4] | 221.1 [144.7 to 337.8] | 258.3 [149.1 to 447.3] | 206.0 [121.1 to 350.6]
  Serotype 18C, Day 30: number analyzed (Participants) | 30 | 30 | 31 | 32
  Serotype 18C, Day 30 | 6975.0 [4497.5 to 10817.4] | 6435.2 [4221.1 to 9810.6] | 6911.0 [4397.8 to 10860.5] | 6405.1 [3931.0 to 10436.3]
  Serotype 19A, Day 1 | 937.2 [507.7 to 1730.0] | 484.6 [298.1 to 787.8] | 581.6 [339.7 to 995.8] | 582.8 [354.0 to 959.6]
  Serotype 19A, Day 30: number analyzed (Participants) | 30 | 30 | 31 | 32
  Serotype 19A, Day 30 | 6568.1 [4520.8 to 9580.6] | 8343.0 [4962.4 to 14026.8] | 8461.9 [5175.4 to 13835.4] | 9721.7 [6666.3 to 14177.5]
  Serotype 19F, Day 1 | 498.4 [263.2 to 943.7] | 477.2 [272.1 to 836.9] | 380.5 [232.2 to 623.3] | 340.1 [192.6 to 600.5]
  Serotype 19F, Day 30: number analyzed (Participants) | 30 | 30 | 31 | 32
  Serotype 19F, Day 30 | 7144.4 [4342.7 to 11753.5] | 9886.9 [7035.8 to 13893.5] | 10142.9 [5870.0 to 17526.0] | 7176.5 [4272.9 to 12053.2]
  Serotype 23F, Day 1 | 254.2 [145.0 to 445.7] | 236.4 [156.9 to 356.4] | 230.0 [122.4 to 432.0] | 251.6 [154.6 to 409.4]
  Serotype 23F, Day 30: number analyzed (Participants) | 30 | 30 | 31 | 32
  Serotype 23F, Day 30 | 5338.2 [3015.8 to 9448.9] | 5759.0 [3467.1 to 9565.8] | 7435.0 [4423.9 to 12495.6] | 11580.6 [6105.4 to 21965.8]
Statistical Analysis 1: Comparison: Stage 1, Group 1 Adults, ASP3772 Low Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 1, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.08, 95% CI 2-sided [0.52 to 2.23]
Statistical Analysis 2: Comparison: Stage 1, Group 1 Adults, ASP3772 Medium Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 1, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.00, 95% CI 2-sided [0.51 to 1.98]
Statistical Analysis 3: Comparison: Stage 1, Group 1 Adults, ASP3772 High Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 1, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.43, 95% CI 2-sided [0.72 to 2.83]
Statistical Analysis 4: Comparison: Stage 1, Group 1 Adults, ASP3772 Low Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 3, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.26, 95% CI 2-sided [0.59 to 2.68]
Statistical Analysis 5: Comparison: Stage 1, Group 1 Adults, ASP3772 Medium Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 3, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.65, 95% CI 2-sided [0.90 to 3.05]
Statistical Analysis 6: Comparison: Stage 1, Group 1 Adults, ASP3772 High Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 3, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.24, 95% CI 2-sided [0.68 to 2.25]
Statistical Analysis 7: Comparison: Stage 1, Group 1 Adults, ASP3772 Low Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 4, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.03, 95% CI 2-sided [0.49 to 2.15]
Statistical Analysis 8: Comparison: Stage 1, Group 1 Adults, ASP3772 Medium Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 4, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 0.82, 95% CI 2-sided [0.39 to 1.74]
Statistical Analysis 9: Comparison: Stage 1, Group 1 Adults, ASP3772 High Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 4, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.24, 95% CI 2-sided [0.59 to 2.59]
Statistical Analysis 10: Comparison: Stage 1, Group 1 Adults, ASP3772 Low Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 5, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.71, 95% CI 2-sided [0.75 to 3.91]
Statistical Analysis 11: Comparison: Stage 1, Group 1 Adults, ASP3772 Medium Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 5, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 0.72, 95% CI 2-sided [0.36 to 1.46]
Statistical Analysis 12: Comparison: Stage 1, Group 1 Adults, ASP3772 High Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 5, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 0.93, 95% CI 2-sided [0.47 to 1.84]
Statistical Analysis 13: Comparison: Stage 1, Group 1 Adults, ASP3772 Low Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 6A, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.19, 95% CI 2-sided [0.57 to 2.52]
Statistical Analysis 14: Comparison: Stage 1, Group 1 Adults, ASP3772 Medium Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 6A, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.28, 95% CI 2-sided [0.64 to 2.56]
Statistical Analysis 15: Comparison: Stage 1, Group 1 Adults, ASP3772 High Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 6A, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.09, 95% CI 2-sided [0.52 to 2.28]
Statistical Analysis 16: Comparison: Stage 1, Group 1 Adults, ASP3772 Low Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 6B, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.23, 95% CI 2-sided [0.49 to 3.09]
Statistical Analysis 17: Comparison: Stage 1, Group 1 Adults, ASP3772 Medium Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 6B, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 0.96, 95% CI 2-sided [0.43 to 2.14]
Statistical Analysis 18: Comparison: Stage 1, Group 1 Adults, ASP3772 High Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 6B, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 0.81, 95% CI 2-sided [0.37 to 1.73]
Statistical Analysis 19: Comparison: Stage 1, Group 1 Adults, ASP3772 Low Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 7F, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.51, 95% CI 2-sided [0.76 to 3.01]
Statistical Analysis 20: Comparison: Stage 1, Group 1 Adults, ASP3772 Medium Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 7F, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.16, 95% CI 2-sided [0.69 to 1.94]
Statistical Analysis 21: Comparison: Stage 1, Group 1 Adults, ASP3772 High Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 7F, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.69, 95% CI 2-sided [0.98 to 2.91]
Statistical Analysis 22: Comparison: Stage 1, Group 1 Adults, ASP3772 Low Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 9V, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.09, 95% CI 2-sided [0.54 to 2.22]
Statistical Analysis 23: Comparison: Stage 1, Group 1 Adults, ASP3772 Medium Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 9V, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 0.74, 95% CI 2-sided [0.41 to 1.36]
Statistical Analysis 24: Comparison: Stage 1, Group 1 Adults, ASP3772 High Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 9V, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 0.85, 95% CI 2-sided [0.47 to 1.55]
Statistical Analysis 25: Comparison: Stage 1, Group 1 Adults, ASP3772 Low Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 14, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 2.05, 95% CI 2-sided [0.84 to 4.99]
Statistical Analysis 26: Comparison: Stage 1, Group 1 Adults, ASP3772 Medium Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 14, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 2.60, 95% CI 2-sided [1.13 to 5.98]
Statistical Analysis 27: Comparison: Stage 1, Group 1 Adults, ASP3772 High Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 14, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 0.89, 95% CI 2-sided [0.37 to 2.15]
Statistical Analysis 28: Comparison: Stage 1, Group 1 Adults, ASP3772 Low Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 18C, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.37, 95% CI 2-sided [0.61 to 3.06]
Statistical Analysis 29: Comparison: Stage 1, Group 1 Adults, ASP3772 Medium Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 18C, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.07, 95% CI 2-sided [0.55 to 2.09]
Statistical Analysis 30: Comparison: Stage 1, Group 1 Adults, ASP3772 High Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 18C, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.25, 95% CI 2-sided [0.59 to 2.65]
Statistical Analysis 31: Comparison: Stage 1, Group 1 Adults, ASP3772 Low Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 19A, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.61, 95% CI 2-sided [0.74 to 3.49]
Statistical Analysis 32: Comparison: Stage 1, Group 1 Adults, ASP3772 Medium Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 19A, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 0.83, 95% CI 2-sided [0.42 to 1.65]
Statistical Analysis 33: Comparison: Stage 1, Group 1 Adults, ASP3772 High Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 19A, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.00, 95% CI 2-sided [0.49 to 2.05]
Statistical Analysis 34: Comparison: Stage 1, Group 1 Adults, ASP3772 Low Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 19F, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.47, 95% CI 2-sided [0.63 to 3.39]
Statistical Analysis 35: Comparison: Stage 1, Group 1 Adults, ASP3772 Medium Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 19F, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.40, 95% CI 2-sided [0.64 to 3.07]
Statistical Analysis 36: Comparison: Stage 1, Group 1 Adults, ASP3772 High Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 19F, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.12, 95% CI 2-sided [0.53 to 2.34]
Statistical Analysis 37: Comparison: Stage 1, Group 1 Adults, ASP3772 Low Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 23F, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.01, 95% CI 2-sided [0.49 to 2.09]
Statistical Analysis 38: Comparison: Stage 1, Group 1 Adults, ASP3772 Medium Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 23F, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 0.94, 95% CI 2-sided [0.50 to 1.75]
Statistical Analysis 39: Comparison: Stage 1, Group 1 Adults, ASP3772 High Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 23F, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 0.91, 95% CI 2-sided [0.42 to 2.00]
Statistical Analysis 40: Comparison: Stage 1, Group 1 Adults, ASP3772 Low Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 1, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 0.70, 95% CI 2-sided [0.38 to 1.29]
Statistical Analysis 41: Comparison: Stage 1, Group 1 Adults, ASP3772 Medium Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 1, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 0.95, 95% CI 2-sided [0.52 to 1.73]
Statistical Analysis 42: Comparison: Stage 1, Group 1 Adults, ASP3772 High Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 1, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.50, 95% CI 2-sided [0.84 to 2.66]
Statistical Analysis 43: Comparison: Stage 1, Group 1 Adults, ASP3772 Low Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 3, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.38, 95% CI 2-sided [0.84 to 2.28]
Statistical Analysis 44: Comparison: Stage 1, Group 1 Adults, ASP3772 Medium Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 3, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 2.68, 95% CI 2-sided [1.71 to 4.19]
Statistical Analysis 45: Comparison: Stage 1, Group 1 Adults, ASP3772 High Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 3, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 3.87, 95% CI 2-sided [2.47 to 6.06]
Statistical Analysis 46: Comparison: Stage 1, Group 1 Adults, ASP3772 Low Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 4, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.27, 95% CI 2-sided [0.70 to 2.30]
Statistical Analysis 47: Comparison: Stage 1, Group 1 Adults, ASP3772 Medium Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 4, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.02, 95% CI 2-sided [0.57 to 1.81]
Statistical Analysis 48: Comparison: Stage 1, Group 1 Adults, ASP3772 High Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 4, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 2.24, 95% CI 2-sided [1.21 to 4.15]
Statistical Analysis 49: Comparison: Stage 1, Group 1 Adults, ASP3772 Low Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 5, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.58, 95% CI 2-sided [0.70 to 3.57]
Statistical Analysis 50: Comparison: Stage 1, Group 1 Adults, ASP3772 Medium Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 5, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 0.84, 95% CI 2-sided [0.35 to 2.05]
Statistical Analysis 51: Comparison: Stage 1, Group 1 Adults, ASP3772 High Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 5, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.49, 95% CI 2-sided [0.65 to 3.39]
Statistical Analysis 52: Comparison: Stage 1, Group 1 Adults, ASP3772 Low Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 6A, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 0.89, 95% CI 2-sided [0.41 to 1.93]
Statistical Analysis 53: Comparison: Stage 1, Group 1 Adults, ASP3772 Medium Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 6A, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 0.77, 95% CI 2-sided [0.33 to 1.79]
Statistical Analysis 54: Comparison: Stage 1, Group 1 Adults, ASP3772 High Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 6A, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 0.69, 95% CI 2-sided [0.32 to 1.48]
Statistical Analysis 55: Comparison: Stage 1, Group 1 Adults, ASP3772 Low Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 6B, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.26, 95% CI 2-sided [0.57 to 2.83]
Statistical Analysis 56: Comparison: Stage 1, Group 1 Adults, ASP3772 Medium Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 6B, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 0.75, 95% CI 2-sided [0.31 to 1.81]
Statistical Analysis 57: Comparison: Stage 1, Group 1 Adults, ASP3772 High Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 6B, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 0.88, 95% CI 2-sided [0.39 to 1.97]
Statistical Analysis 58: Comparison: Stage 1, Group 1 Adults, ASP3772 Low Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 7F, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.86, 95% CI 2-sided [1.05 to 3.30]
Statistical Analysis 59: Comparison: Stage 1, Group 1 Adults, ASP3772 Medium Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 7F, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.98, 95% CI 2-sided [1.10 to 3.55]
Statistical Analysis 60: Comparison: Stage 1, Group 1 Adults, ASP3772 High Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 7F, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 2.88, 95% CI 2-sided [1.62 to 5.12]
Statistical Analysis 61: Comparison: Stage 1, Group 1 Adults, ASP3772 Low Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 9V, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 0.96, 95% CI 2-sided [0.49 to 1.87]
Statistical Analysis 62: Comparison: Stage 1, Group 1 Adults, ASP3772 Medium Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 9V, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.39, 95% CI 2-sided [0.74 to 2.62]
Statistical Analysis 63: Comparison: Stage 1, Group 1 Adults, ASP3772 High Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 9V, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.68, 95% CI 2-sided [0.87 to 3.27]
Statistical Analysis 64: Comparison: Stage 1, Group 1 Adults, ASP3772 Low Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 14, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.01, 95% CI 2-sided [0.41 to 2.53]
Statistical Analysis 65: Comparison: Stage 1, Group 1 Adults, ASP3772 Medium Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 14, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.08, 95% CI 2-sided [0.45 to 2.60]
Statistical Analysis 66: Comparison: Stage 1, Group 1 Adults, ASP3772 High Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 14, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 2.09, 95% CI 2-sided [0.86 to 5.04]
Statistical Analysis 67: Comparison: Stage 1, Group 1 Adults, ASP3772 Low Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 18C, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.09, 95% CI 2-sided [0.57 to 2.07]
Statistical Analysis 68: Comparison: Stage 1, Group 1 Adults, ASP3772 Medium Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 18C, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.00, 95% CI 2-sided [0.53 to 1.89]
Statistical Analysis 69: Comparison: Stage 1, Group 1 Adults, ASP3772 High Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 18C, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.08, 95% CI 2-sided [0.56 to 2.07]
Statistical Analysis 70: Comparison: Stage 1, Group 1 Adults, ASP3772 Low Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 19A, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 0.68, 95% CI 2-sided [0.40 to 1.14]
Statistical Analysis 71: Comparison: Stage 1, Group 1 Adults, ASP3772 Medium Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 19A, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 0.86, 95% CI 2-sided [0.46 to 1.61]
Statistical Analysis 72: Comparison: Stage 1, Group 1 Adults, ASP3772 High Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 19A, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 0.87, 95% CI 2-sided [0.47 to 1.60]
Statistical Analysis 73: Comparison: Stage 1, Group 1 Adults, ASP3772 Low Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 19F, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.00, 95% CI 2-sided [0.49 to 2.01]
Statistical Analysis 74: Comparison: Stage 1, Group 1 Adults, ASP3772 Medium Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 19F, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.38, 95% CI 2-sided [0.75 to 2.53]
Statistical Analysis 75: Comparison: Stage 1, Group 1 Adults, ASP3772 High Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 19F, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.41, 95% CI 2-sided [0.68 to 2.96]
Statistical Analysis 76: Comparison: Stage 1, Group 1 Adults, ASP3772 Low Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 23F, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 0.46, 95% CI 2-sided [0.20 to 1.07]
Statistical Analysis 77: Comparison: Stage 1, Group 1 Adults, ASP3772 Medium Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 23F, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 0.50, 95% CI 2-sided [0.22 to 1.11]
Statistical Analysis 78: Comparison: Stage 1, Group 1 Adults, ASP3772 High Dose vs Stage 1, Group 1, PCV13 Pooled Comparator; Serotype 23F, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 0.64, 95% CI 2-sided [0.29 to 1.44]

16. Secondary Outcome: Geometric Mean Fold Rise (GMFR) for Unique Serotypes IgG [Stage 1, Group 1]
Description: Immunological responses were assessed in terms of IgG GMFRs. The assessed serotypes were: 2, 8, 9N, 10A, 11A, 12F, 15B, 17F, 20B, 22F, and 33F.
Time Frame: At Day 30
Population: The analysis was performed on the Full Analysis Set which consisted of all randomized participants who received a vaccination in this study with either ASP3772 or PCV13, had at least 1 postvaccination measurement and for whom immunogenicity data was collected for specific serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Stage 1, Group 1 Adults, ASP3772 Low Dose | Stage 1, Group 1 Adults, ASP3772 Medium Dose | Stage 1, Group 1 Adults, ASP3772 High Dose | Stage 1, Group 1, PCV13 Pooled Comparator
Number analyzed (Participants) | 30 | 30 | 32 | 32
fold rise
  Serotype 2: number analyzed (Participants) | 30 | 30 | 31 | 32
  Serotype 2 | 29.7 [18.1 to 49.0] | 34.5 [19.7 to 60.4] | 66.5 [40.3 to 109.6] | 1.2 [1.1 to 1.3]
  Serotype 8: number analyzed (Participants) | 30 | 30 | 31 | 32
  Serotype 8 | 35.8 [20.3 to 63.4] | 57.7 [34.6 to 96.2] | 102.7 [62.2 to 169.5] | 1.3 [1.0 to 1.7]
  Serotype 9N: number analyzed (Participants) | 30 | 30 | 31 | 32
  Serotype 9N | 32.3 [19.8 to 52.6] | 39.5 [23.6 to 66.1] | 51.6 [29.0 to 91.7] | 3.5 [2.4 to 5.0]
  Serotype 10A: number analyzed (Participants) | 30 | 30 | 31 | 32
  Serotype 10A | 14.8 [9.7 to 22.6] | 10.0 [6.6 to 15.0] | 16.2 [10.9 to 24.2] | 1.7 [1.3 to 2.3]
  Serotype 11A: number analyzed (Participants) | 30 | 30 | 31 | 32
  Serotype 11A | 6.8 [3.9 to 11.9] | 11.2 [6.4 to 19.6] | 22.3 [15.1 to 33.2] | 1.1 [1.0 to 1.1]
  Serotype 12F: number analyzed (Participants) | 30 | 30 | 31 | 32
  Serotype 12F | 17.1 [10.7 to 27.5] | 30.6 [19.5 to 47.9] | 31.7 [20.1 to 50.2] | 1.5 [1.2 to 2.0]
  Serotype 15B: number analyzed (Participants) | 30 | 30 | 31 | 32
  Serotype 15B | 16.0 [8.4 to 30.5] | 18.7 [10.8 to 32.3] | 32.2 [17.6 to 58.8] | 1.5 [1.1 to 2.0]
  Serotype 17F: number analyzed (Participants) | 30 | 30 | 31 | 32
  Serotype 17F | 28.2 [16.5 to 48.2] | 48.0 [32.6 to 70.7] | 70.4 [41.2 to 120.4] | 1.2 [1.1 to 1.4]
  Serotype 20B: number analyzed (Participants) | 30 | 30 | 31 | 32
  Serotype 20B | 7.2 [5.0 to 10.5] | 11.4 [8.5 to 15.4] | 12.7 [8.3 to 19.6] | 1.1 [1.0 to 1.3]
  Serotype 22F: number analyzed (Participants) | 30 | 30 | 31 | 32
  Serotype 22F | 30.4 [15.7 to 59.0] | 60.7 [30.2 to 122.0] | 52.6 [23.2 to 119.4] | 1.1 [1.1 to 1.2]
  Serotype 33F: number analyzed (Participants) | 30 | 30 | 31 | 32
  Serotype 33F | 17.6 [11.8 to 26.2] | 37.9 [25.7 to 55.7] | 25.5 [16.8 to 38.8] | 2.2 [1.7 to 2.9]

17. Secondary Outcome: Percentage of Participants With Unique Serotypes IgG of Greater Than or Equal to (>=) 4-fold Increase, [Stage 1, Group 1]
Description: Immunological responses were assessed in terms of percentage of participants with serotype-specific IgG concentration >=4-fold increase. The assessed serotypes were: 2, 8, 9N, 10A, 11A, 12F, 15B, 17F, 20B, 22F, 33F.
Time Frame: At Day 30
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Stage 1, Group 1 Adults, ASP3772 Low Dose | Stage 1, Group 1 Adults, ASP3772 Medium Dose | Stage 1, Group 1 Adults, ASP3772 High Dose | Stage 1, Group 1, PCV13 Pooled Comparator
Number analyzed (Participants) | 30 | 31 | 31 | 32
Percentage of participants
  Serotype 2: number analyzed (Participants) | 30 | 30 | 31 | 32
  Serotype 2 | 93.3 [77.9 to 99.2] | 86.7 [69.3 to 96.2] | 96.8 [83.3 to 99.9] | 0 [0.0 to 10.9]
  Serotype 8: number analyzed (Participants) | 30 | 30 | 31 | 32
  Serotype 8 | 93.3 [77.9 to 99.2] | 96.7 [82.8 to 99.9] | 96.8 [83.3 to 99.9] | 3.1 [0.1 to 16.2]
  Serotype 9N: number analyzed (Participants) | 30 | 30 | 31 | 32
  Serotype 9N | 93.3 [77.9 to 99.2] | 90.0 [73.5 to 97.9] | 90.3 [74.2 to 98.0] | 43.8 [26.4 to 62.3]
  Serotype 10A | 90.0 [73.5 to 97.9] | 83.3 [65.3 to 94.4] | 90.3 [74.2 to 98.0] | 18.8 [7.2 to 36.4]
  Serotype 11A: number analyzed (Participants) | 30 | 30 | 31 | 32
  Serotype 11A | 56.7 [37.4 to 74.5] | 70.0 [50.6 to 85.3] | 96.8 [83.3 to 99.9] | 0 [0.0 to 10.9]
  Serotype 12F: number analyzed (Participants) | 30 | 30 | 31 | 32
  Serotype 12F | 90.0 [73.5 to 97.9] | 93.3 [77.9 to 99.2] | 96.8 [83.3 to 99.9] | 6.3 [0.8 to 20.8]
  Serotype 15B: number analyzed (Participants) | 30 | 30 | 31 | 32
  Serotype 15B | 76.7 [57.7 to 90.1] | 80.0 [61.4 to 92.3] | 87.1 [70.2 to 96.4] | 3.1 [0.1 to 16.2]
  Serotype 17F: number analyzed (Participants) | 30 | 30 | 31 | 32
  Serotype 17F | 90.0 [73.5 to 97.9] | 100.0 [88.4 to 100.0] | 93.5 [78.6 to 99.2] | 3.1 [0.1 to 16.2]
  Serotype 20B: number analyzed (Participants) | 30 | 30 | 31 | 32
  Serotype 20B | 70.0 [50.6 to 85.3] | 86.7 [69.3 to 96.2] | 83.9 [66.3 to 94.5] | 0 [0.0 to 10.9]
  Serotype 22F: number analyzed (Participants) | 30 | 30 | 31 | 32
  Serotype 22F | 86.7 [69.3 to 96.2] | 93.3 [77.9 to 99.2] | 80.6 [62.5 to 92.5] | 0 [0.0 to 10.9]
  Serotype 33F: number analyzed (Participants) | 30 | 30 | 31 | 32
  Serotype 33F | 90.0 [73.5 to 97.9] | 100.0 [88.4 to 100.0] | 96.8 [83.3 to 99.9] | 21.9 [9.3 to 40.0]

18. Secondary Outcome: GMTs for Unique Serotype OPA Titer, [Stage 1, Group 1]
Description: Immunological responses were assessed in terms of OPA GMTs. The assessed serotypes were: 2, 8, 9N, 10A, 11A, 12F, 15B, 17F, 20B, 22F, 33F.
Time Frame: At Day 30
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Stage 1, Group 1 Adults, ASP3772 Low Dose | Stage 1, Group 1 Adults, ASP3772 Medium Dose | Stage 1, Group 1 Adults, ASP3772 High Dose | Stage 1, Group 1, PCV13 Pooled Comparator
Number analyzed (Participants) | 29 | 29 | 31 | 31
Titers
  Serotype 2: number analyzed (Participants) | 28 | 29 | 31 | 31
  Serotype 2 | 5702.0 [4352.7 to 7469.6] | 5966.2 [4328.1 to 8224.2] | 6963.2 [5705.4 to 8498.1] | 177.9 [70.8 to 447.1]
  Serotype 8 | 2122.5 [1542.8 to 2920.0] | 2000.8 [1408.2 to 2842.8] | 3254.8 [2465.2 to 4297.1] | 37.0 [17.5 to 78.4]
  Serotype 9N: number analyzed (Participants) | 28 | 29 | 31 | 31
  Serotype 9N | 8525.4 [6424.8 to 11312.7] | 10826.3 [6622.7 to 17698.1] | 10215.2 [7413.7 to 14075.3] | 2856.4 [1941.7 to 4202.0]
  Serotype 10A: number analyzed (Participants) | 29 | 29 | 29 | 29
  Serotype 10A | 5542.2 [3611.7 to 8504.6] | 6094.6 [3267.7 to 11367.1] | 7764.2 [5609.5 to 10746.5] | 189.7 [59.3 to 606.7]
  Serotype 11A: number analyzed (Participants) | 25 | 27 | 28 | 29
  Serotype 11A | 2020.9 [1398.4 to 2920.4] | 2034.8 [1459.3 to 2837.3] | 3195.5 [2446.0 to 4174.7] | 244.3 [100.5 to 594.0]
  Serotype 12F: number analyzed (Participants) | 29 | 28 | 28 | 23
  Serotype 12F | 5536.4 [3663.1 to 8367.7] | 6501.7 [4629.6 to 9130.9] | 6630.9 [5206.3 to 8445.2] | 358.7 [155.3 to 828.5]
  Serotype 15B: number analyzed (Participants) | 28 | 26 | 28 | 25
  Serotype 15B | 17128.6 [9415.4 to 31160.9] | 15042.0 [8201.1 to 27589.4] | 21608.2 [12903.6 to 36184.7] | 2497.2 [1303.0 to 4785.7]
  Serotype 17F: number analyzed (Participants) | 29 | 29 | 30 | 29
  Serotype 17F | 15011.7 [9861.1 to 22852.3] | 10352.1 [7518.3 to 14253.9] | 18396.7 [12958.7 to 26116.8] | 388.6 [138.0 to 1094.5]
  Serotype 20B: number analyzed (Participants) | 28 | 28 | 29 | 30
  Serotype 20B | 17250.5 [11193.0 to 26586.3] | 37410.1 [24523.3 to 57068.9] | 36949.9 [25705.3 to 53113.4] | 1828.6 [969.2 to 3450.3]
  Serotype 22F: number analyzed (Participants) | 28 | 24 | 27 | 21
  Serotype 22F | 6897.2 [4411.0 to 10784.6] | 9221.2 [5497.3 to 15467.6] | 7085.5 [4866.3 to 10316.7] | 628.2 [213.8 to 1846.2]
  Serotype 33F: number analyzed (Participants) | 29 | 28 | 28 | 29
  Serotype 33F | 13291.8 [9855.6 to 17926.0] | 16419.1 [11478.7 to 23485.7] | 21934.8 [13531.7 to 35556.0] | 647.7 [257.1 to 1631.7]

19. Secondary Outcome: GMTs for Serotype-specific OPA Titer, [Stage 2, Group 2]
Description: Immunological responses were assessed in terms of OPA GMTs and expressed as titers. The assessed serotypes were: 1, 3,4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F.
Time Frame: At Day 1 and Day 30
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Stage 2, Group 2 Older Adults, ASP3772 Low Dose | Stage 2, Group 2 Older Adults, ASP3772 Medium Dose | Stage 2, Group 2 Older Adults, ASP3772 High Dose | Stage 2, Group 2, PCV13 Pooled Comparator
Number analyzed (Participants) | 98 | 105 | 85 | 94
Titers
  Serotype 1, Day 1: number analyzed (Participants) | 97 | 85 | 66 | 87
  Serotype 1, Day 1 | 8.7 [7.0 to 10.8] | 15.0 [10.6 to 21.2] | 7.9 [6.2 to 10.1] | 10.8 [8.2 to 14.3]
  Serotype 1, Day 30: number analyzed (Participants) | 98 | 102 | 83 | 94
  Serotype 1, Day 30 | 158.0 [109.7 to 227.5] | 165.0 [115.0 to 236.8] | 242.0 [173.6 to 337.3] | 189.3 [122.6 to 292.4]
  Serotype 3, Day 1: number analyzed (Participants) | 90 | 80 | 64 | 77
  Serotype 3, Day 1 | 17.6 [12.6 to 24.4] | 19.0 [13.4 to 27.0] | 12.5 [8.9 to 17.5] | 13.2 [9.6 to 18.0]
  Serotype 3, Day 30: number analyzed (Participants) | 88 | 92 | 68 | 79
  Serotype 3, Day 30 | 276.8 [212.9 to 359.9] | 390.5 [318.1 to 479.3] | 480.4 [378.0 to 610.6] | 153.0 [117.2 to 199.9]
  Serotype 4, Day 1: number analyzed (Participants) | 94 | 84 | 63 | 81
  Serotype 4, Day 1 | 14.5 [10.1 to 20.8] | 19.6 [13.5 to 28.4] | 12.6 [8.7 to 18.3] | 18.0 [11.8 to 27.4]
  Serotype 4, Day 30: number analyzed (Participants) | 95 | 102 | 84 | 91
  Serotype 4, Day 30 | 718.9 [525.5 to 983.3] | 691.5 [536.5 to 891.3] | 903.6 [685.2 to 1191.5] | 732.9 [492.8 to 1090.1]
  Serotype 5, Day 1: number analyzed (Participants) | 95 | 85 | 68 | 86
  Serotype 5, Day 1 | 12.8 [8.8 to 18.7] | 17.2 [11.5 to 25.7] | 11.4 [7.6 to 17.2] | 13.0 [8.9 to 19.0]
  Serotype 5, Day 30: number analyzed (Participants) | 96 | 104 | 85 | 92
  Serotype 5, Day 30 | 394.6 [269.4 to 578.1] | 456.1 [329.9 to 630.4] | 678.9 [477.7 to 964.7] | 315.1 [206.5 to 480.8]
  Serotype 6A, Day 1: number analyzed (Participants) | 93 | 81 | 62 | 79
  Serotype 6A, Day 1 | 30.6 [20.8 to 44.8] | 51.8 [32.4 to 82.9] | 51.1 [30.8 to 85.0] | 31.7 [20.4 to 49.4]
  Serotype 6A, Day 30: number analyzed (Participants) | 80 | 96 | 79 | 84
  Serotype 6A, Day 30 | 1409.7 [961.9 to 2065.9] | 1834.9 [1366.6 to 2463.6] | 1900.5 [1285.5 to 2809.7] | 2045.8 [1342.3 to 3118.1]
  Serotype 6B, Day 1: number analyzed (Participants) | 86 | 84 | 59 | 77
  Serotype 6B, Day 1 | 79.1 [50.6 to 123.8] | 82.6 [52.3 to 130.4] | 84.3 [50.0 to 142.0] | 71.6 [43.8 to 117.1]
  Serotype 6B, Day 30: number analyzed (Participants) | 95 | 104 | 83 | 93
  Serotype 6B, Day 30 | 2194.2 [1552.9 to 3100.4] | 1978.5 [1510.8 to 2591.0] | 1941.6 [1433.5 to 2629.7] | 2324.0 [1686.0 to 3203.5]
  Serotype 7F, Day 1: number analyzed (Participants) | 81 | 77 | 57 | 79
  Serotype 7F, Day 1 | 91.7 [54.2 to 155.2] | 146.6 [87.0 to 247.2] | 112.0 [59.5 to 210.9] | 108.7 [62.6 to 188.8]
  Serotype 7F, Day 30: number analyzed (Participants) | 91 | 99 | 72 | 85
  Serotype 7F, Day 30 | 2631.4 [2067.9 to 3348.5] | 2742.0 [2218.9 to 3388.4] | 3230.9 [2440.3 to 4277.6] | 3084.0 [2461.6 to 3863.9]
  Serotype 9V, Day 1: number analyzed (Participants) | 84 | 71 | 58 | 72
  Serotype 9V, Day 1 | 80.7 [50.2 to 129.7] | 96.6 [56.7 to 164.5] | 82.0 [44.1 to 152.8] | 123.7 [73.0 to 209.6]
  Serotype 9V, Day 30: number analyzed (Participants) | 84 | 94 | 71 | 80
  Serotype 9V, Day 30 | 1715.4 [1183.3 to 2486.6] | 1453.7 [1090.8 to 1937.3] | 2503.0 [1887.8 to 3318.8] | 2060.2 [1402.9 to 3025.5]
  Serotype 14, Day 1: number analyzed (Participants) | 95 | 83 | 67 | 84
  Serotype 14, Day 1 | 85.8 [55.5 to 132.6] | 153.6 [95.2 to 247.8] | 186.7 [115.9 to 300.8] | 141.2 [84.7 to 235.6]
  Serotype 14, Day 30: number analyzed (Participants) | 96 | 104 | 84 | 93
  Serotype 14, Day 30 | 1912.6 [1411.8 to 2591.2] | 1273.4 [917.5 to 1767.2] | 2221.0 [1594.0 to 3094.7] | 1437.7 [1009.8 to 2046.8]
  Serotype 18C, Day 1: number analyzed (Participants) | 94 | 77 | 67 | 83
  Serotype 18C, Day 1 | 38.3 [26.2 to 56.0] | 98.2 [62.0 to 155.5] | 41.2 [27.6 to 61.5] | 71.4 [46.3 to 110.2]
  Serotype 18C, Day 30: number analyzed (Participants) | 90 | 101 | 81 | 85
  Serotype 18C, Day 30 | 1325.5 [973.0 to 1805.7] | 1461.3 [1121.2 to 1904.6] | 1951.6 [1434.1 to 2655.9] | 1483.9 [1028.2 to 2141.5]
  Serotype 19A, Day 1: number analyzed (Participants) | 96 | 84 | 68 | 83
  Serotype 19A, Day 1 | 128.2 [87.7 to 187.4] | 193.2 [131.2 to 284.4] | 141.4 [93.5 to 213.9] | 167.7 [112.1 to 250.8]
  Serotype 19A, Day 30: number analyzed (Participants) | 97 | 105 | 81 | 90
  Serotype 19A, Day 30 | 2062.6 [1635.1 to 2602.0] | 2081.5 [1665.4 to 2601.6] | 2417.8 [1810.4 to 3229.0] | 2115.0 [1652.4 to 2707.1]
  Serotype 19F, Day 1: number analyzed (Participants) | 89 | 76 | 63 | 79
  Serotype 19F, Day 1 | 79.1 [54.0 to 115.7] | 84.7 [55.8 to 128.4] | 62.3 [41.1 to 94.6] | 100.6 [65.9 to 153.6]
  Serotype 19F, Day 30: number analyzed (Participants) | 90 | 101 | 82 | 89
  Serotype 19F, Day 30 | 1672.1 [1260.2 to 2218.6] | 1626.9 [1307.5 to 2024.3] | 2295.5 [1706.7 to 3087.3] | 1102.6 [798.0 to 1523.3]
  Serotype 23F, Day 1: number analyzed (Participants) | 91 | 83 | 58 | 82
  Serotype 23F, Day 1 | 26.0 [17.2 to 39.3] | 32.0 [20.8 to 49.1] | 27.8 [17.6 to 43.8] | 23.4 [16.0 to 34.3]
  Serotype 23F, Day 30: number analyzed (Participants) | 91 | 98 | 73 | 83
  Serotype 23F, Day 30 | 537.4 [355.1 to 813.3] | 567.0 [413.3 to 777.8] | 722.2 [462.0 to 1128.7] | 800.1 [494.7 to 1294.1]
Statistical Analysis 1: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 1, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.80, 95% CI 2-sided [0.56 to 1.14]
Statistical Analysis 2: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 1, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.39, 95% CI 2-sided [0.89 to 2.16]
Statistical Analysis 3: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 1, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.73, 95% CI 2-sided [0.51 to 1.06]
Statistical Analysis 4: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 3, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.33, 95% CI 2-sided [0.85 to 2.09]
Statistical Analysis 5: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 3, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.45, 95% CI 2-sided [0.91 to 2.30]
Statistical Analysis 6: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 3, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.95, 95% CI 2-sided [0.60 to 1.49]
Statistical Analysis 7: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 4, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.81, 95% CI 2-sided [0.46 to 1.40]
Statistical Analysis 8: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 4, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.09, 95% CI 2-sided [0.62 to 1.91]
Statistical Analysis 9: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 4, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.70, 95% CI 2-sided [0.40 to 1.23]
Statistical Analysis 10: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 5, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.98, 95% CI 2-sided [0.58 to 1.68]
Statistical Analysis 11: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 5, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.32, 95% CI 2-sided [0.76 to 2.29]
Statistical Analysis 12: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 5, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.88, 95% CI 2-sided [0.51 to 1.53]
Statistical Analysis 13: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 6A, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.96, 95% CI 2-sided [0.54 to 1.72]
Statistical Analysis 14: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 6B, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.10, 95% CI 2-sided [0.57 to 2.14]
Statistical Analysis 15: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 6A, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.63, 95% CI 2-sided [0.86 to 3.10]
Statistical Analysis 16: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 6A, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.61, 95% CI 2-sided [0.83 to 3.14]
Statistical Analysis 17: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 6B, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.15, 95% CI 2-sided [0.59 to 2.24]
Statistical Analysis 18: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 6B, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.18, 95% CI 2-sided [0.58 to 2.39]
Statistical Analysis 19: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 7F, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.84, 95% CI 2-sided [0.40 to 1.80]
Statistical Analysis 20: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 7F, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.35, 95% CI 2-sided [0.63 to 2.87]
Statistical Analysis 21: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 7F, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.03, 95% CI 2-sided [0.45 to 2.37]
Statistical Analysis 22: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 9V, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.65, 95% CI [0.32 to 1.32]
Statistical Analysis 23: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 9V, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.78, 95% CI 2-sided [0.37 to 1.64]
Statistical Analysis 24: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 9V, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.66, 95% CI 2-sided [0.30 to 1.49]
Statistical Analysis 25: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 14, Day 1; Test type: Other; t-test, 1 sided; Ratio of GMT = 0.61, 95% CI 2-sided [0.31 to 1.18]
Statistical Analysis 26: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 14, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.09, 95% CI 2-sided [0.54 to 2.18]
Statistical Analysis 27: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 14, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.32, 95% CI 2-sided [0.66 to 2.65]
Statistical Analysis 28: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 18C, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.54, 95% CI 2-sided [0.30 to 0.95]
Statistical Analysis 29: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 18C, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.37, 95% CI 2-sided [0.73 to 2.57]
Statistical Analysis 30: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 18C, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.58, 95% CI 2-sided [0.32 to 1.04]
Statistical Analysis 31: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 19A, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.76, 95% CI 2-sided [0.44 to 1.32]
Statistical Analysis 32: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 19A, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.15, 95% CI 2-sided [0.66 to 2.01]
Statistical Analysis 33: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 19A, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.84, 95% CI 2-sided [0.48 to 1.50]
Statistical Analysis 34: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 19F, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.79, 95% CI 2-sided [0.45 to 1.38]
Statistical Analysis 35: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 19F, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.84, 95% CI 2-sided [0.47 to 1.52]
Statistical Analysis 36: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 19F, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.62, 95% CI 2-sided [0.34 to 1.12]
Statistical Analysis 37: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 23F, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.11, 95% CI 2-sided [0.64 to 1.94]
Statistical Analysis 38: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 23F, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.37, 95% CI 2-sided [0.77 to 2.42]
Statistical Analysis 39: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 23F, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.19, 95% CI 2-sided [0.66 to 2.14]
Statistical Analysis 40: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 1, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.83, 95% CI 2-sided [0.47 to 1.47]
Statistical Analysis 41: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 1, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.87, 95% CI 2-sided [0.50 to 1.53]
Statistical Analysis 42: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 1, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.28, 95% CI 2-sided [0.74 to 2.20]
Statistical Analysis 43: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 2, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 25.03, 95% CI 2-sided [16.33 to 38.34]
Statistical Analysis 44: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 2, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 21.99, 95% CI 2-sided [14.31 to 33.77]
Statistical Analysis 45: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 2, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 35.38, 95% CI 2-sided [23.09 to 54.22]
Statistical Analysis 46: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 3, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.81, 95% CI 2-sided [1.25 to 2.62]
Statistical Analysis 47: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 3, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 2.55, 95% CI 2-sided [1.83 to 3.56]
Statistical Analysis 48: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 3, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 3.14, 95% CI 2-sided [2.20 to 4.48]
Statistical Analysis 49: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 4, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.98, 95% CI 2-sided [0.59 to 1.62]
Statistical Analysis 50: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 4, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.94, 95% CI 2-sided [0.59 to 1.51]
Statistical Analysis 51: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 4, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.23, 95% CI 2-sided [0.76 to 1.99]
Statistical Analysis 52: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 5, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.25, 95% CI 2-sided [0.71 to 2.21]
Statistical Analysis 53: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 5, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.45, 95% CI 2-sided [0.85 to 2.46]
Statistical Analysis 54: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 5, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 2.15, 95% CI 2-sided [1.25 to 3.72]
Statistical Analysis 55: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 6B, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.94, 95% CI 2-sided [0.59 to 1.51]
Statistical Analysis 56: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 6B, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.85, 95% CI 2-sided [0.56 to 1.29]
Statistical Analysis 57: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 6B, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.84, 95% CI 2-sided [0.54 to 1.30]
Statistical Analysis 58: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 7F, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.85, 95% CI 2-sided [0.61 to 1.18]
Statistical Analysis 59: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 7F, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.89, 95% CI 2-sided [0.65 to 1.21]
Statistical Analysis 60: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 7F, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.05, 95% CI 2-sided [0.73 to 1.50]
Statistical Analysis 61: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 8, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 19.46, 95% CI 2-sided [12.26 to 30.87]
Statistical Analysis 62: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 8, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 19.65, 95% CI 2-sided [12.07 to 32.00]
Statistical Analysis 63: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 8, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 41.87, 95% CI 2-sided [26.20 to 66.90]
Statistical Analysis 64: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 9N, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 4.75, 95% CI 2-sided [3.06 to 7.36]
Statistical Analysis 65: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 9N, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 5.66, 95% CI 2-sided [3.83 to 8.37]
Statistical Analysis 66: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 9N, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 7.84, 95% CI 2-sided [5.19 to 11.82]
Statistical Analysis 67: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 9V, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.83, 95% CI 2-sided [0.49 to 1.42]
Statistical Analysis 68: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 9V, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.71, 95% CI 2-sided [0.44 to 1.14]
Statistical Analysis 69: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 9V, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.21, 95% CI 2-sided [0.76 to 1.95]
Statistical Analysis 70: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 6A, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.69, 95% CI 2-sided [0.39 to 1.21]
Statistical Analysis 71: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 6A, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.90, 95% CI 2-sided [0.54 to 1.50]
Statistical Analysis 72: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 6A, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.93, 95% CI 2-sided [0.53 to 1.64]
Statistical Analysis 73: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 14, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.33, 95% CI 2-sided [0.84 to 2.11]
Statistical Analysis 74: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 14, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.89, 95% CI 2-sided [0.55 to 1.43]
Statistical Analysis 75: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 14, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.54, 95% CI 2-sided [0.95 to 2.50]
Statistical Analysis 76: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 18C, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.89, 95% CI 2-sided [0.55 to 1.44]
Statistical Analysis 77: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 18C, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.98, 95% CI 2-sided [0.63 to 1.54]
Statistical Analysis 78: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 18C, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.32, 95% CI 2-sided [0.82 to 2.12]
Statistical Analysis 79: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 19A, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.98, 95% CI 2-sided [0.70 to 1.37]
Statistical Analysis 80: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 19A, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.98, 95% CI 2-sided [0.71 to 1.37]
Statistical Analysis 81: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 19A, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.14, 95% CI 2-sided [0.78 to 1.67]
Statistical Analysis 82: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 19F, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.52, 95% CI [0.99 to 2.32]
Statistical Analysis 83: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 19F, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.48, 95% CI 2-sided [1.00 to 2.18]
Statistical Analysis 84: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 19F, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 2.08, 95% CI 2-sided [1.35 to 3.22]
Statistical Analysis 85: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 23F, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.67, 95% CI 2-sided [0.36 to 1.26]
Statistical Analysis 86: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 23F, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.71, 95% CI 2-sided [0.40 to 1.26]
Statistical Analysis 87: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 23F, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.90, 95% CI 2-sided [0.47 to 1.73]

20. Secondary Outcome: GMCs for Serotype-specific IgG, [Stage 2, Group 2]
Description: as for outcome 15
Time Frame: At Day 1 and Day 30
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Stage 2, Group 2 Older Adults, ASP3772 Low Dose | Stage 2, Group 2 Older Adults, ASP3772 Medium Dose | Stage 2, Group 2 Older Adults, ASP3772 High Dose | Stage 2, Group 2, PCV13 Pooled Comparator
Number analyzed (Participants) | 98 | 106 | 86 | 96
Titers
  Serotype 1, Day 1: number analyzed (Participants) | 97 | 87 | 70 | 88
  Serotype 1, Day 1 | 268.1 [199.7 to 359.9] | 551.9 [382.2 to 796.9] | 263.0 [178.6 to 387.3] | 297.6 [208.9 to 424.0]
  Serotype 1, Day 30 | 4510.3 [3281.4 to 6199.3] | 5730.2 [4361.3 to 7528.7] | 6436.8 [4867.6 to 8511.8] | 5510.9 [3954.4 to 7680.1]
  Serotype 3, Day 1: number analyzed (Participants) | 97 | 87 | 70 | 88
  Serotype 3, Day 1 | 76.0 [57.7 to 100.1] | 109.0 [80.7 to 147.3] | 65.4 [46.4 to 92.1] | 60.8 [45.2 to 81.7]
  Serotype 3, Day 30 | 846.4 [643.4 to 1113.4] | 1348.7 [1097.3 to 1657.8] | 1657.6 [1289.6 to 2130.5] | 409.5 [316.1 to 530.6]
  Serotype 4, Day 1: number analyzed (Participants) | 97 | 87 | 70 | 88
  Serotype 4, Day 1 | 128.1 [99.9 to 164.3] | 183.9 [134.7 to 250.9] | 105.6 [82.0 to 136.0] | 158.6 [114.7 to 219.4]
  Serotype 4, Day 30 | 1518.9 [1090.2 to 2116.4] | 1866.0 [1447.4 to 2405.5] | 2013.4 [1485.8 to 2728.3] | 1923.5 [1365.7 to 2709.3]
  Serotype 5, Day 1: number analyzed (Participants) | 97 | 87 | 70 | 88
  Serotype 5, Day 1 | 175.6 [121.8 to 253.2] | 258.6 [178.7 to 374.3] | 163.1 [107.0 to 248.4] | 162.9 [114.8 to 231.1]
  Serotype 5, Day 30 | 3261.2 [2256.5 to 4713.2] | 3236.7 [2383.4 to 4395.6] | 4752.5 [3244.3 to 6961.8] | 2490.5 [1627.7 to 3810.6]
  Serotype 6A, Day 1: number analyzed (Participants) | 97 | 87 | 70 | 88
  Serotype 6A, Day 1 | 172.0 [118.0 to 250.9] | 270.9 [187.5 to 391.5] | 273.4 [176.4 to 423.9] | 195.6 [137.4 to 278.4]
  Serotype 6A, Day 30 | 3132.7 [2122.1 to 4624.6] | 3850.7 [2866.6 to 5172.5] | 4438.5 [3016.6 to 6530.8] | 3640.4 [2464.8 to 5376.9]
  Serotype 6B, Day 1: number analyzed (Participants) | 97 | 87 | 70 | 88
  Serotype 6B, Day 1 | 162.7 [112.3 to 235.9] | 291.3 [193.1 to 439.4] | 221.4 [140.6 to 348.5] | 139.1 [94.4 to 205.0]
  Serotype 6B, Day 30 | 2835.9 [1906.8 to 4217.9] | 4135.1 [2913.0 to 5870.0] | 5088.3 [3384.8 to 7649.1] | 2869.5 [1900.3 to 4333.0]
  Serotype 7F, Day 1: number analyzed (Participants) | 97 | 87 | 70 | 88
  Serotype 7F, Day 1 | 279.9 [202.1 to 387.6] | 438.6 [301.8 to 637.3] | 250.3 [156.7 to 399.8] | 276.8 [190.8 to 401.4]
  Serotype 7F, Day 30 | 5660.9 [4186.2 to 7655.1] | 5710.7 [4401.8 to 7408.8] | 6123.2 [4437.8 to 8448.6] | 3684.2 [2801.5 to 4845.0]
  Serotype 9V, Day 1: number analyzed (Participants) | 97 | 87 | 70 | 88
  Serotype 9V, Day 1 | 183.6 [139.7 to 241.4] | 364.5 [255.1 to 520.9] | 229.1 [158.9 to 330.4] | 232.6 [167.5 to 322.9]
  Serotype 9V, Day 30 | 2990.4 [2221.0 to 4026.3] | 3798.3 [2917.8 to 4944.5] | 5006.8 [3701.4 to 6772.5] | 2316.5 [1601.7 to 3350.4]
  Serotype 14, Day 1: number analyzed (Participants) | 97 | 87 | 70 | 88
  Serotype 14, Day 1 | 732.5 [490.1 to 1095.0] | 1329.0 [877.6 to 2012.6] | 867.2 [553.0 to 1360.0] | 997.3 [639.0 to 1556.6]
  Serotype 14, Day 30 | 7024.7 [4809.3 to 10260.8] | 8927.8 [6494.0 to 12273.7] | 11822.1 [8177.6 to 17090.8] | 7087.9 [4885.3 to 10283.5]
  Serotype 18C, Day 1: number analyzed (Participants) | 97 | 87 | 70 | 88
  Serotype 18C, Day 1 | 313.5 [225.5 to 435.8] | 695.1 [483.0 to 1000.3] | 354.1 [228.9 to 547.6] | 454.9 [315.5 to 655.9]
  Serotype 18C, Day 30 | 3647.5 [2598.6 to 5119.8] | 6242.2 [4764.7 to 8177.8] | 6189.4 [4553.9 to 8412.3] | 6012.3 [4479.0 to 8070.6]
  Serotype 19A, Day 1: number analyzed (Participants) | 97 | 87 | 70 | 88
  Serotype 19A, Day 1 | 710.7 [533.1 to 947.5] | 1157.8 [820.2 to 1634.4] | 906.3 [641.7 to 1279.8] | 867.1 [634.2 to 1185.7]
  Serotype 19A, Day 30 | 7704.4 [5669.3 to 10469.9] | 9838.0 [7745.0 to 12496.7] | 11047.0 [7767.0 to 15712.0] | 9233.5 [7068.3 to 12061.9]
  Serotype 19F, Day 1: number analyzed (Participants) | 97 | 87 | 70 | 88
  Serotype 19F, Day 1 | 357.9 [252.7 to 506.7] | 542.8 [373.9 to 787.9] | 424.9 [276.6 to 652.4] | 429.9 [299.8 to 616.4]
  Serotype 19F, Day 30 | 5479.0 [3926.5 to 7645.2] | 7737.1 [5853.8 to 10226.3] | 10186.4 [7337.3 to 14141.8] | 4568.2 [3313.7 to 6297.6]
  Serotype 23F, Day 1: number analyzed (Participants) | 97 | 87 | 70 | 88
  Serotype 23F, Day 1 | 190.8 [131.4 to 276.9] | 210.7 [142.5 to 311.6] | 210.7 [136.7 to 324.7] | 176.5 [118.7 to 262.3]
  Serotype 23F, Day 30 | 2569.9 [1806.9 to 3655.1] | 2480.7 [1907.8 to 3225.7] | 3535.7 [2495.3 to 5010.0] | 2989.8 [1984.3 to 4504.8]
Statistical Analysis 1: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 1, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 0.90, 95% CI 2-sided [0.57 to 1.42]
Statistical Analysis 2: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 1, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.85, 95% CI 2-sided [1.12 to 3.08]
Statistical Analysis 3: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 1, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 0.88, 95% CI 2-sided [0.53 to 1.49]
Statistical Analysis 4: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 3, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.25, 95% CI 2-sided [0.84 to 1.87]
Statistical Analysis 5: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 3, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.79, 95% CI 2-sided [1.18 to 2.73]
Statistical Analysis 6: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 3, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.08, 95% CI 2-sided [0.69 to 1.69]
Statistical Analysis 7: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 4, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 0.81, 95% CI 2-sided [0.54 to 1.21]
Statistical Analysis 8: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 4, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.16, 95% CI 2-sided [0.74 to 1.81]
Statistical Analysis 9: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 4, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 0.67, 95% CI 2-sided [0.44 to 1.00]
Statistical Analysis 10: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 5, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.08, 95% CI 2-sided [0.65 to 1.78]
Statistical Analysis 11: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 5, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.59, 95% CI 2-sided [0.96 to 2.63]
Statistical Analysis 12: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 5, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.00, 95% CI 2-sided [0.58 to 1.72]
Statistical Analysis 13: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 6A, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 0.88, 95% CI 2-sided [0.53 to 1.47]
Statistical Analysis 14: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 6A, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.39, 95% CI 2-sided [0.83 to 2.30]
Statistical Analysis 15: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 6A, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.40, 95% CI 2-sided [0.80 to 2.44]
Statistical Analysis 16: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 6B, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.17, 95% CI 2-sided [0.69 to 1.99]
Statistical Analysis 17: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 6B, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 2.09, 95% CI 2-sided [1.19 to 3.67]
Statistical Analysis 18: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 6B, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.59, 95% CI 2-sided [0.88 to 2.88]
Statistical Analysis 19: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 7F, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.01, 95% CI 2-sided [0.62 to 1.65]
Statistical Analysis 20: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 7F, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.58, 95% CI 2-sided [0.94 to 2.67]
Statistical Analysis 21: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 7F, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 0.90, 95% CI 2-sided [0.50 to 1.64]
Statistical Analysis 22: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 9V, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 0.79, 95% CI 2-sided [0.52 to 1.21]
Statistical Analysis 23: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 9V, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.57, 95% CI 2-sided [0.97 to 2.54]
Statistical Analysis 24: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 9V, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 0.99, 95% CI 2-sided [0.60 to 1.60]
Statistical Analysis 25: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 14, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 0.73, 95% CI 2-sided [0.40 to 1.33]
Statistical Analysis 26: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 14, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.33, 95% CI 2-sided [0.73 to 2.44]
Statistical Analysis 27: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 14, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 0.87, 95% CI 2-sided [0.46 to 1.63]
Statistical Analysis 28: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 18C, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 0.69, 95% CI 2-sided [0.42 to 1.12]
Statistical Analysis 29: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 18C, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.53, 95% CI 2-sided [0.92 to 2.55]
Statistical Analysis 30: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 18C, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 0.78, 95% CI 2-sided [0.44 to 1.37]
Statistical Analysis 31: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 19A, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 0.82, 95% CI 2-sided [0.54 to 1.25]
Statistical Analysis 32: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 19A, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.34, 95% CI 2-sided [0.84 to 2.12]
Statistical Analysis 33: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 19A, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.05, 95% CI 2-sided [0.66 to 1.66]
Statistical Analysis 34: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 19F, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 0.83, 95% CI 2-sided [0.51 to 1.37]
Statistical Analysis 35: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 19F, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.26, 95% CI 2-sided [0.75 to 2.11]
Statistical Analysis 36: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 19F, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 0.99, 95% CI 2-sided [0.57 to 1.72]
Statistical Analysis 37: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 23F, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.08, 95% CI 2-sided [0.63 to 1.86]
Statistical Analysis 38: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 23F, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.19, 95% CI 2-sided [0.69 to 2.08]
Statistical Analysis 39: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 23F, Day 1; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.19, 95% CI 2-sided [0.67 to 2.14]
Statistical Analysis 40: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 1, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 0.82, 95% CI 2-sided [0.52 to 1.29]
Statistical Analysis 41: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 1, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.04, 95% CI 2-sided [0.68 to 1.59]
Statistical Analysis 42: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 1, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.17, 95% CI 2-sided [0.76 to 1.80]
Statistical Analysis 43: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 3, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 2.07, 95% CI 2-sided [1.42 to 3.01]
Statistical Analysis 44: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 3, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 3.29, 95% CI 2-sided [2.37 to 4.58]
Statistical Analysis 45: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 3, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 4.05, 95% CI 2-sided [2.83 to 5.79]
Statistical Analysis 46: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 4, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 0.79, 95% CI 2-sided [0.49 to 1.27]
Statistical Analysis 47: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 4, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 0.97, 95% CI 2-sided [0.63 to 1.48]
Statistical Analysis 48: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 4, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.05, 95% CI 2-sided [0.66 to 1.65]
Statistical Analysis 49: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 5, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.31, 95% CI 2-sided [0.75 to 2.29]
Statistical Analysis 50: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 5, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.30, 95% CI 2-sided [0.77 to 2.19]
Statistical Analysis 51: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 5, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.91, 95% CI 2-sided [1.08 to 3.37]
Statistical Analysis 52: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 6A, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 0.86, 95% CI 2-sided [0.50 to 1.49]
Statistical Analysis 53: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 6A, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.06, 95% CI 2-sided [0.65 to 1.72]
Statistical Analysis 54: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 6A, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.22, 95% CI 2-sided [0.71 to 2.10]
Statistical Analysis 55: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 6B, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 0.99, 95% CI 2-sided [0.56 to 1.75]
Statistical Analysis 56: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 6B, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.44, 95% CI 2-sided [0.84 to 2.47]
Statistical Analysis 57: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 6B, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.77, 95% CI 2-sided [1.00 to 3.15]
Statistical Analysis 58: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 7F, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.54, 95% CI 2-sided [1.02 to 2.30]
Statistical Analysis 59: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 7F, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.55, 95% CI 2-sided [1.06 to 2.26]
Statistical Analysis 60: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 7F, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.66, 95% CI 2-sided [1.09 to 2.53]
Statistical Analysis 61: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 9V, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.29, 95% CI 2-sided [0.81 to 2.07]
Statistical Analysis 62: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 9V, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.64, 95% CI 2-sided [1.04 to 2.57]
Statistical Analysis 63: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 9V, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 2.16, 95% CI 2-sided [1.35 to 3.47]
Statistical Analysis 64: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 14, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 0.99, 95% CI 2-sided [0.58 to 1.68]
Statistical Analysis 65: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 14, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.26, 95% CI 2-sided [0.77 to 2.05]
Statistical Analysis 66: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 14, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.67, 95% CI 2-sided [0.99 to 2.81]
Statistical Analysis 67: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 18C, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 0.61, 95% CI 2-sided [0.39 to 0.95]
Statistical Analysis 68: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 18C, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.04, 95% CI 2-sided [0.70 to 1.54]
Statistical Analysis 69: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 18C, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.03, 95% CI 2-sided [0.67 to 1.57]
Statistical Analysis 70: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 19A, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 0.83, 95% CI 2-sided [0.56 to 1.25]
Statistical Analysis 71: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 19A, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.07, 95% CI 2-sided [0.75 to 1.52]
Statistical Analysis 72: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 19A, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.20, 95% CI 2-sided [0.77 to 1.86]
Statistical Analysis 73: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 19F, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.20, 95% CI 2-sided [0.76 to 1.90]
Statistical Analysis 74: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 19F, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.69, 95% CI 2-sided [1.11 to 2.58]
Statistical Analysis 75: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 19F, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 2.23, 95% CI 2-sided [1.41 to 3.52]
Statistical Analysis 76: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 23F, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 0.86, 95% CI 2-sided [0.50 to 1.47]
Statistical Analysis 77: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 23F, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 0.83, 95% CI 2-sided [0.51 to 1.35]
Statistical Analysis 78: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 2, PCV13 Pooled Comparator; Serotype 23F, Day 30; Test type: Other; t-test, 2 sided; Ratio of GMC = 1.18, 95% CI 2-sided [0.69 to 2.02]

21. Secondary Outcome: GMFR for Unique Serotypes IgG, [Stage 2, Group 2]
Description: as for outcome 16
Time Frame: At Day 30
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Stage 2, Group 2 Older Adults, ASP3772 Low Dose | Stage 2, Group 2 Older Adults, ASP3772 Medium Dose | Stage 2, Group 2 Older Adults, ASP3772 High Dose | Stage 2, Group 2, PCV13 Pooled Comparator
Number analyzed (Participants) | 95 | 87 | 70 | 88
fold rise
  Serotype 2 | 17.0 [12.4 to 23.5] | 12.2 [8.5 to 17.5] | 22.6 [15.7 to 32.6] | 1.0 [1.0 to 1.1]
  Serotype 8 | 24.4 [17.5 to 34.0] | 18.0 [12.3 to 26.3] | 45.7 [30.4 to 68.6] | 1.2 [1.0 to 1.3]
  Serotype 9N | 19.5 [14.1 to 27.0] | 12.4 [8.6 to 17.8] | 32.0 [22.6 to 45.4] | 2.3 [1.9 to 2.8]
  Serotype 10A | 13.9 [10.7 to 18.1] | 11.9 [8.7 to 16.4] | 19.3 [13.7 to 27.1] | 1.1 [1.0 to 1.2]
  Serotype 11A | 10.5 [7.9 to 14.0] | 9.9 [7.2 to 13.7] | 18.2 [12.8 to 25.9] | 1.1 [1.0 to 1.2]
  Serotype 12F | 10.6 [7.7 to 14.6] | 11.6 [8.2 to 16.3] | 14.4 [9.7 to 21.5] | 1.1 [1.0 to 1.1]
  Serotype 15B | 13.0 [9.6 to 17.5] | 9.6 [6.8 to 13.6] | 20.3 [13.5 to 30.5] | 1.8 [1.4 to 2.4]
  Serotype 17F | 26.4 [19.5 to 35.6] | 17.1 [12.3 to 23.9] | 27.2 [18.8 to 39.4] | 1.1 [1.0 to 1.1]
  Serotype 20B | 10.1 [8.0 to 12.9] | 10.4 [7.7 to 13.9] | 15.6 [11.8 to 20.8] | 1.1 [1.0 to 1.1]
  Serotype 22F | 20.5 [14.6 to 28.6] | 16.2 [11.2 to 23.3] | 30.5 [20.9 to 44.7] | 1.1 [1.0 to 1.2]
  Serotype 33F | 12.2 [9.1 to 16.5] | 10.5 [7.5 to 14.7] | 16.7 [11.6 to 24.0] | 1.1 [1.0 to 1.1]

22. Secondary Outcome: Percentage of Participants With Unique Serotype-specific IgG Concentration of Greater Than or Equal to (>=) 4-fold Increase, [Stage 2, Group 2]
Description: Immunological responses were assessed in terms of percentage of participants with unique serotypes IgG concentration >=4-fold increase. The assessed serotypes were: 2, 8, 9N, 10A, 11A, 12F, 15B, 17F, 20B, 22F, 33F.
Time Frame: At Day 30
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Stage 2, Group 2 Older Adults, ASP3772 Low Dose | Stage 2, Group 2 Older Adults, ASP3772 Medium Dose | Stage 2, Group 2 Older Adults, ASP3772 High Dose | Stage 2, Group 2, PCV13 Pooled Comparator
Number analyzed (Participants) | 95 | 87 | 70 | 88
Percentage of participants
  Serotype 2 | 77.9 [68.2 to 85.8] | 67.8 [56.9 to 77.4] | 81.4 [70.3 to 89.7] | 1.1 [0.0 to 6.2]
  Serotype 8 | 85.3 [76.5 to 91.7] | 75.9 [65.5 to 84.4] | 87.1 [77.0 to 93.9] | 2.3 [0.3 to 8.0]
  Serotype 9N | 84.2 [75.3 to 90.9] | 66.7 [55.7 to 76.4] | 87.1 [77.0 to 93.9] | 25.0 [16.4 to 35.4]
  Serotype 10A | 82.1 [72.9 to 89.2] | 74.7 [64.3 to 83.4] | 85.7 [75.3 to 92.9] | 1.1 [0.0 to 6.2]
  Serotype 11A | 72.6 [62.5 to 81.3] | 67.8 [56.9 to 77.4] | 84.3 [73.6 to 91.9] | 0 [0.0 to 4.1]
  Serotype 12F | 66.3 [55.9 to 75.7] | 72.4 [61.8 to 81.5] | 71.4 [59.4 to 81.6] | 0 [0.0 to 4.1]
  Serotype 15B | 72.6 [62.5 to 81.3] | 65.5 [54.6 to 75.4] | 74.3 [62.4 to 84.0] | 17.0 [9.9 to 26.6]
  Serotype 17F | 92.6 [85.4 to 97.0] | 82.8 [73.2 to 90.0] | 90.0 [80.5 to 95.9] | 0 [0.0 to 4.1]
  Serotype 20B | 81.1 [71.7 to 88.4] | 74.7 [64.3 to 83.4] | 84.3 [73.6 to 91.9] | 1.1 [0.0 to 6.2]
  Serotype 22F | 82.1 [72.9 to 89.2] | 71.3 [60.6 to 80.5] | 90.0 [80.5 to 95.9] | 1.1 [0.0 to 6.2]
  Serotype 33F | 75.8 [65.9 to 84.0] | 66.7 [55.7 to 76.4] | 80.0 [68.7 to 88.6] | 0 [0.0 to 4.1]

23. Secondary Outcome: Dose Response in OPA Titer for ASP3772 (Stage 2, Group 2)
Description: An analysis of covariance (ANCOVA) model was conducted with age categories (65 to 74 years and 75 to 85 years) serving as covariates, and treatment groups (ASP3772 1 µg, 2 µg, and 5 µg) as the factor of interest. The natural logarithm (log) of pneumococcal OPA titers for each serotype were examined to assess the dose-response relationship. The assessed serotypes were: 1, 2, 3, 4, 5, 6A, 6B, 7F, 8, 9N, 9V, 10A, 11A, 12F, 14, 15B, 17F, 18C, 19A, 19F,20B, 22F, 23F, and 33F. he assessed serotypes were: 1, 2, 3, 4, 5, 6A, 6B, 7F, 8, 9N, 9V, 10A, 11A, 12F, 14, 15B, 17F, 18C, 19A, 19F,20B, 22F, 23F, and 33F.
Time Frame: At Day 30
Population: The analysis was performed on the Full Analysis Set which consisted of all randomized participants who received a vaccination in this study with ASP3772, had at least 1 post vaccination measurement and for whom immunogenicity data was collected for specific serotype.
Measure: Least Squares Mean (95% Confidence Interval); unit: ln(titers)
Arm/Group | Stage 2, Group 2 Older Adults, ASP3772 Low Dose | Stage 2, Group 2 Older Adults, ASP3772 Medium Dose | Stage 2, Group 2 Older Adults, ASP3772 High Dose
Number analyzed (Participants) | 98 | 105 | 85
ln(titers)
  Serotype 1, Day 30: number analyzed (Participants) | 98 | 102 | 83
  Serotype 1, Day 30 | 5.0 [4.5 to 5.4] | 5.0 [4.6 to 5.4] | 5.4 [4.9 to 5.8]
  Serotype 2, Day 30: number analyzed (Participants) | 96 | 105 | 84
  Serotype 2, Day 30 | 7.0 [6.8 to 7.3] | 6.9 [6.7 to 7.2] | 7.4 [7.1 to 7.6]
  Serotype 3, Day 30: number analyzed (Participants) | 88 | 92 | 68
  Serotype 3, Day 30 | 5.6 [5.4 to 5.9] | 6.0 [5.7 to 6.2] | 6.2 [5.9 to 6.5]
  Serotype 4, Day 30: number analyzed (Participants) | 95 | 102 | 84
  Serotype 4, Day 30 | 6.3 [6.0 to 6.6] | 6.3 [6.0 to 6.6] | 6.5 [6.2 to 6.9]
  Serotype 5, Day 30: number analyzed (Participants) | 96 | 104 | 85
  Serotype 5, Day 30 | 6.1 [5.7 to 6.6] | 6.3 [5.9 to 6.7] | 6.7 [6.2 to 7.1]
  Serotype 6A, Day 30: number analyzed (Participants) | 80 | 96 | 79
  Serotype 6A, Day 30 | 7.2 [6.7 to 7.6] | 7.4 [7.0 to 7.8] | 7.5 [7.0 to 7.9]
  Serotype 6B, Day 30: number analyzed (Participants) | 95 | 104 | 83
  Serotype 6B, Day 30 | 7.6 [7.2 to 8.0] | 7.5 [7.2 to 7.9] | 7.5 [7.1 to 7.9]
  Serotype 7F, Day 30: number analyzed (Participants) | 91 | 99 | 72
  Serotype 7F, Day 30 | 7.7 [7.4 to 7.9] | 7.7 [7.5 to 8.0] | 7.9 [7.6 to 8.2]
  Serotype 8, Day 30: number analyzed (Participants) | 96 | 104 | 79
  Serotype 8, Day 30 | 7.0 [6.7 to 7.3] | 7.0 [6.7 to 7.3] | 7.8 [7.4 to 8.1]
  Serotype 9N, Day 30: number analyzed (Participants) | 97 | 100 | 80
  Serotype 9N, Day 30 | 7.8 [7.5 to 8.1] | 8.0 [7.8 to 8.3] | 8.3 [8.0 to 8.6]
  Serotype 9V, Day 30: number analyzed (Participants) | 84 | 94 | 71
  Serotype 9V, Day 30 | 7.5 [7.1 to 7.8] | 7.3 [6.9 to 7.6] | 7.8 [7.4 to 8.2]
  Serotype 10A, Day 30: number analyzed (Participants) | 97 | 102 | 80
  Serotype 10A, Day 30 | 7.4 [7.0 to 7.8] | 7.7 [7.3 to 8.1] | 7.8 [7.4 to 8.3]
  Serotype 11A, Day 30: number analyzed (Participants) | 96 | 102 | 81
  Serotype 11A, Day 30 | 5.8 [5.5 to 6.2] | 6.1 [5.8 to 6.4] | 6.6 [6.2 to 6.9]
  Serotype 12F, Day 30: number analyzed (Participants) | 95 | 102 | 82
  Serotype 12F, Day 30 | 7.0 [6.6 to 7.5] | 6.8 [6.4 to 7.2] | 7.3 [6.8 to 7.7]
  Serotype 14, Day 30: number analyzed (Participants) | 96 | 104 | 84
  Serotype 14, Day 30 | 7.3 [6.9 to 7.7] | 7.0 [6.6 to 7.3] | 7.5 [7.1 to 7.9]
  Serotype 15B, Day 30: number analyzed (Participants) | 88 | 86 | 72
  Serotype 15B, Day 30 | 8.5 [8.1 to 8.8] | 8.2 [7.9 to 8.5] | 8.6 [8.2 to 9.0]
  Serotype 17F, Day 30: number analyzed (Participants) | 97 | 103 | 81
  Serotype 17F, Day 30 | 8.0 [7.8 to 8.3] | 7.9 [7.6 to 8.2] | 8.3 [8.0 to 8.6]
  Serotype 18C, Day 30: number analyzed (Participants) | 90 | 101 | 81
  Serotype 18C, Day 30 | 6.9 [6.5 to 7.2] | 7.0 [6.7 to 7.3] | 7.3 [6.9 to 7.6]
  Serotype 19A, Day 30: number analyzed (Participants) | 97 | 105 | 81
  Serotype 19A, Day 30 | 7.4 [7.1 to 7.7] | 7.4 [7.2 to 7.7] | 7.6 [7.2 to 7.9]
  Serotype 19F, Day 30: number analyzed (Participants) | 90 | 101 | 82
  Serotype 19F, Day 30 | 7.2 [6.9 to 7.6] | 7.2 [6.9 to 7.5] | 7.6 [7.2 to 7.9]
  Serotype 20B, Day 30: number analyzed (Participants) | 92 | 95 | 73
  Serotype 20B, Day 30 | 9.4 [9.0 to 9.8] | 9.2 [8.8 to 9.6] | 9.8 [9.4 to 10.2]
  Serotype 22F, Day 30: number analyzed (Participants) | 93 | 93 | 81
  Serotype 22F, Day 30 | 7.4 [7.1 to 7.7] | 7.3 [7.0 to 7.6] | 7.6 [7.2 to 7.9]
  Serotype 23F, Day 30: number analyzed (Participants) | 91 | 98 | 73
  Serotype 23F, Day 30 | 6.4 [5.9 to 6.9] | 6.4 [6.0 to 6.9] | 6.7 [6.2 to 7.2]
  Serotype 33F, Day 30: number analyzed (Participants) | 95 | 101 | 83
  Serotype 33F, Day 30 | 8.4 [8.1 to 8.8] | 8.4 [8.1 to 8.7] | 8.6 [8.3 to 9.0]
Statistical Analysis 1: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 Medium Dose; Serotype 1, Day 30; Test type: Other; p = 0.805, ANCOVA; Mean Difference = 0.1, 95% CI 2-sided [-0.4 to 0.5]
Statistical Analysis 2: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 1, Day 30; Test type: Other; p = 0.102, ANCOVA; Mean Difference = 0.4, 95% CI 2-sided [-0.1 to 0.9]
Statistical Analysis 3: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 1, Day 30; Test type: Other; p = 0.158, ANCOVA; Mean Difference = 0.4, 95% CI 2-sided [-0.1 to 0.9]
Statistical Analysis 4: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 Medium Dose; Serotype 2, Day 30; Test type: Other; p = 0.596, ANCOVA; Mean Difference = -0.1, 95% CI 2-sided [-0.4 to 0.2]
Statistical Analysis 5: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 2, Day 30; Test type: Other; p = 0.025, ANCOVA; Mean Difference = 0.3, 95% CI 2-sided [0.0 to 0.7]
Statistical Analysis 6: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 2, Day 30; Test type: Other; p = 0.005, ANCOVA; Mean Difference = 0.4, 95% CI 2-sided [0.1 to 0.7]
Statistical Analysis 7: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 Medium Dose; Serotype 3, Day 30; Test type: Other; p = 0.037, ANCOVA; Mean Difference = 0.3, 95% CI 2-sided [0.0 to 0.7]
Statistical Analysis 8: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 3, Day 30; Test type: Other; p = 0.002, ANCOVA; Mean Difference = 0.6, 95% CI 2-sided [0.2 to 0.9]
Statistical Analysis 9: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 3, Day 30; Test type: Other; p = 0.230, ANCOVA; Mean Difference = 0.2, 95% CI 2-sided [-0.1 to 0.6]
Statistical Analysis 10: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 Medium Dose; Serotype 4, Day 30; Test type: Other; p = 0.984, ANCOVA; Mean Difference = 0.0, 95% CI 2-sided [-0.4 to 0.4]
Statistical Analysis 11: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 4, Day 30; Test type: Other; p = 0.262, ANCOVA; Mean Difference = 0.2, 95% CI 2-sided [-0.2 to 0.6]
Statistical Analysis 12: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 4, Day 30; Test type: Other; p = 0.264, ANCOVA; Mean Difference = 0.2, 95% CI 2-sided [-0.2 to 0.6]
Statistical Analysis 13: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 Medium Dose; Serotype 5, Day 30; Test type: Other; p = 0.638, ANCOVA; Mean Difference = 0.1, 95% CI 2-sided [-0.4 to 0.6]
Statistical Analysis 14: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 5, Day 30; Test type: Other; p = 0.036, ANCOVA; Mean Difference = 0.5, 95% CI 2-sided [0.0 to 1.0]
Statistical Analysis 15: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 5, Day 30; Test type: Other; p = 0.094, ANCOVA; Mean Difference = 0.4, 95% CI 2-sided [-0.1 to 0.9]
Statistical Analysis 16: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 Medium Dose; Serotype 6A, Day 30; Test type: Other; p = 0.266, ANCOVA; Mean Difference = 0.3, 95% CI 2-sided [-0.2 to 0.8]
Statistical Analysis 17: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 6A, Day 30; Test type: Other; p = 0.250, ANCOVA; Mean Difference = 0.3, 95% CI 2-sided [-0.2 to 0.8]
Statistical Analysis 18: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 6A, Day 30; Test type: Other; p = 0.927, ANCOVA; Mean Difference = 0.0, 95% CI 2-sided [-0.5 to 0.5]
Statistical Analysis 19: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 Medium Dose; Serotype 6B, Day 30; Test type: Other; p = 0.679, ANCOVA; Mean Difference = -0.1, 95% CI 2-sided [-0.5 to 0.3]
Statistical Analysis 20: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 6B, Day 30; Test type: Other; p = 0.589, ANCOVA; Mean Difference = -0.1, 95% CI 2-sided [-0.6 to 0.3]
Statistical Analysis 21: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 6B, Day 30; Test type: Other; p = 0.880, ANCOVA; Mean Difference = 0.0, 95% CI 2-sided [-0.5 to 0.4]
Statistical Analysis 22: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 Medium Dose; Serotype 7F, Day 30; Test type: Other; p = 0.623, ANCOVA; Mean Difference = 0.1, 95% CI 2-sided [-0.2 to 0.4]
Statistical Analysis 23: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 7F, Day 30; Test type: Other; p = 0.232, ANCOVA; Mean Difference = 0.2, 95% CI 2-sided [-0.1 to 0.6]
Statistical Analysis 24: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 7F, Day 30; Test type: Other; p = 0.451, ANCOVA; Mean Difference = 0.1, 95% CI 2-sided [-0.2 to 0.5]
Statistical Analysis 25: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 Medium Dose; Serotype 8, Day 30; Test type: Other; p = 0.785, ANCOVA; Mean Difference = 0.0, 95% CI 2-sided [-0.3 to 0.4]
Statistical Analysis 26: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 8, Day 30; Test type: Other; p < .001, ANCOVA; Mean Difference = 0.8, 95% CI 2-sided [0.4 to 1.1]
Statistical Analysis 27: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 8, Day 30; Test type: Other; p < .001, ANCOVA; Mean Difference = 0.7, 95% CI 2-sided [0.4 to 1.1]
Statistical Analysis 28: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 Medium Dose; Serotype 9N, Day 30; Test type: Other; p = 0.146, ANCOVA; Mean Difference = 0.2, 95% CI 2-sided [-0.1 to 0.5]
Statistical Analysis 29: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 9N, Day 30; Test type: Other; p = 0.003, ANCOVA; Mean Difference = 0.5, 95% CI 2-sided [0.2 to 0.8]
Statistical Analysis 30: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 9N, Day 30; Test type: Other; p = 0.113, ANCOVA; Mean Difference = 0.3, 95% CI 2-sided [-0.1 to 0.6]
Statistical Analysis 31: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 Medium Dose; Serotype 9V, Day 30; Test type: Other; p = 0.453, ANCOVA; Mean Difference = -0.2, 95% CI 2-sided [-0.6 to 0.3]
Statistical Analysis 32: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 9V, Day 30; Test type: Other; p = 0.111, ANCOVA; Mean Difference = 0.4, 95% CI 2-sided [-0.1 to 0.8]
Statistical Analysis 33: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 9V, Day 30; Test type: Other; p = 0.020, ANCOVA; Mean Difference = 0.5, 95% CI 2-sided [0.1 to 1.0]
Statistical Analysis 34: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 Medium Dose; Serotype 10A, Day 30; Test type: Other; p = 0.218, ANCOVA; Mean Difference = 0.3, 95% CI 2-sided [-0.2 to 0.8]
Statistical Analysis 35: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 10A, Day 30; Test type: Other; p = 0.125, ANCOVA; Mean Difference = 0.4, 95% CI 2-sided [-0.1 to 0.9]
Statistical Analysis 36: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 10A, Day 30; Test type: Other; p = 0.706, ANCOVA; Mean Difference = 0.1, 95% CI 2-sided [-0.4 to 0.6]
Statistical Analysis 37: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 Medium Dose; Serotype 11A, Day 30; Test type: Other; p = 0.246, ANCOVA; Mean Difference = 0.2, 95% CI 2-sided [-0.1 to 0.6]
Statistical Analysis 38: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 11A, Day 30; Test type: Other; p < .001, ANCOVA; Mean Difference = 0.7, 95% CI 2-sided [0.3 to 1.1]
Statistical Analysis 39: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 11A, Day 30; Test type: Other; p = 0.010, ANCOVA; Mean Difference = 0.5, 95% CI 2-sided [0.1 to 0.9]
Statistical Analysis 40: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 Medium Dose; Serotype 12F, Day 30; Test type: Other; p = 0.260, ANCOVA; Mean Difference = -0.3, 95% CI 2-sided [-0.7 to 0.2]
Statistical Analysis 41: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 12F, Day 30; Test type: Other; p = 0.366, ANCOVA; Mean Difference = 0.2, 95% CI 2-sided [-0.3 to 0.7]
Statistical Analysis 42: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 12F, Day 30; Test type: Other; p = 0.046, ANCOVA; Mean Difference = 0.5, 95% CI 2-sided [0.0 to 1.0]
Statistical Analysis 43: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 Medium Dose; Serotype 14, Day 30; Test type: Other; p = 0.101, ANCOVA; Mean Difference = -0.4, 95% CI 2-sided [-0.8 to 0.1]
Statistical Analysis 44: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 14, Day 30; Test type: Other; p = 0.522, ANCOVA; Mean Difference = 0.2, 95% CI [-0.3 to 0.6]
Statistical Analysis 45: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 14, Day 30; Test type: Other; p = 0.026, ANCOVA; Mean Difference = 0.5, 95% CI 2-sided [0.1 to 1.0]
Statistical Analysis 46: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 Medium Dose; Serotype 15B, Day 30; Test type: Other; p = 0.236, ANCOVA; Mean Difference = -0.2, 95% CI 2-sided [-0.6 to 0.2]
Statistical Analysis 47: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 15B, Day 30; Test type: Other; p = 0.528, ANCOVA; Mean Difference = 0.1, 95% CI 2-sided [-0.3 to 0.5]
Statistical Analysis 48: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 15B, Day 30; Test type: Other; p = 0.081, ANCOVA; Mean Difference = 0.4, 95% CI 2-sided [0.0 to 0.8]
Statistical Analysis 49: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 Medium Dose; Serotype 17F, Day 30; Test type: Other; p = 0.388, ANCOVA; Mean Difference = -0.1, 95% CI 2-sided [-0.5 to 0.2]
Statistical Analysis 50: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 17F, Day 30; Test type: Other; p = 0.151, ANCOVA; Mean Difference = 0.3, 95% CI 2-sided [-0.1 to 0.6]
Statistical Analysis 51: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 17F, Day 30; Test type: Other; p = 0.024, ANCOVA; Mean Difference = 0.4, 95% CI 2-sided [0.1 to 0.7]
Statistical Analysis 52: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 Medium Dose; Serotype 18C, Day 30; Test type: Other; p = 0.476, ANCOVA; Mean Difference = 0.1, 95% CI 2-sided [-0.3 to 0.5]
Statistical Analysis 53: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 18C, Day 30; Test type: Other; p = 0.077, ANCOVA; Mean Difference = 0.4, 95% CI 2-sided [0.0 to 0.8]
Statistical Analysis 54: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 18C, Day 30; Test type: Other; p = 0.262, ANCOVA; Mean Difference = 0.2, 95% CI 2-sided [-0.2 to 0.6]
Statistical Analysis 55: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 Medium Dose; Serotype 19A, Day 30; Test type: Other; p = 0.767, ANCOVA; Mean Difference = 0.0, 95% CI 2-sided [-0.3 to 0.4]
Statistical Analysis 56: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 19A, Day 30; Test type: Other; p = 0.364, ANCOVA; Mean Difference = 0.2, 95% CI 2-sided [-0.2 to 0.5]
Statistical Analysis 57: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 19A, Day 30; Test type: Other; p = 0.522, ANCOVA; Mean Difference = 0.1, 95% CI 2-sided [-0.2 to 0.5]
Statistical Analysis 58: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 Medium Dose; Serotype 19F, Day 30; Test type: Other; p = 0.962, ANCOVA; Mean Difference = 0.0, 95% CI 2-sided [-0.4 to 0.4]
Statistical Analysis 59: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 19F, Day 30; Test type: Other; p = 0.091, ANCOVA; Mean Difference = 0.3, 95% CI 2-sided [-0.1 to 0.7]
Statistical Analysis 60: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 19F, Day 30; Test type: Other; p = 0.093, ANCOVA; Mean Difference = 0.3, 95% CI 2-sided [-0.1 to 0.7]
Statistical Analysis 61: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 Medium Dose; Serotype 20B, Day 30; Test type: Other; p = 0.455, ANCOVA; Mean Difference = -0.2, 95% CI 2-sided [-0.6 to 0.3]
Statistical Analysis 62: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 20B, Day 30; Test type: Other; p = 0.093, ANCOVA; Mean Difference = 0.4, 95% CI 2-sided [-0.1 to 0.9]
Statistical Analysis 63: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 20B, Day 30; Test type: Other; p = 0.017, ANCOVA; Mean Difference = 0.6, 95% CI 2-sided [0.1 to 1.1]
Statistical Analysis 64: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 Medium Dose; Serotype 22F, Day 30; Test type: Other; p = 0.561, ANCOVA; Mean Difference = -0.1, 95% CI 2-sided [-0.5 to 0.3]
Statistical Analysis 65: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 22F, Day 30; Test type: Other; p = 0.343, ANCOVA; Mean Difference = 0.2, 95% CI 2-sided [-0.2 to 0.6]
Statistical Analysis 66: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 22F, Day 30; Test type: Other; p = 0.132, ANCOVA; Mean Difference = 0.3, 95% CI 2-sided [-0.1 to 0.7]
Statistical Analysis 67: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 Medium Dose; Serotype 23F, Day 30; Test type: Other; p = 0.898, ANCOVA; Mean Difference = 0.0, 95% CI 2-sided [-0.5 to 0.6]
Statistical Analysis 68: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 23F, Day 30; Test type: Other; p = 0.313, ANCOVA; Mean Difference = 0.3, 95% CI 2-sided [-0.3 to 0.9]
Statistical Analysis 69: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 23F, Day 30; Test type: Other; p = 0.366, ANCOVA; Mean Difference = 0.3, 95% CI 2-sided [-0.3 to 0.8]
Statistical Analysis 70: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 Medium Dose; Serotype 33F, Day 30; Test type: Other; p = 0.961, ANCOVA; Mean Difference = 0.0, 95% CI 2-sided [-0.4 to 0.4]
Statistical Analysis 71: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 33F, Day 30; Test type: Other; p = 0.269, ANCOVA; Mean Difference = 0.2, 95% CI 2-sided [-0.2 to 0.6]
Statistical Analysis 72: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 33F, Day 30; Test type: Other; p = 0.245, ANCOVA; Mean Difference = 0.2, 95% CI 2-sided [-0.2 to 0.6]

24. Secondary Outcome: Dose Response in the IgG Concentrations for ASP3772 [Stage 2, Group 2]
Description: An analysis of covariance (ANCOVA) model was conducted with age categories (65 to 74 years and 75 to 85 years) serving as covariates, and treatment groups (ASP3772 1 µg, 2 µg, and 5 µg) as the factor of interest. The natural logarithm (log) of IgG concentrations for each serotype were examined to assess the dose-response relationship.
Time Frame: At Day 30
Population: as for outcome 23
Measure: Least Squares Mean (95% Confidence Interval); unit: ln(titers)
Arm/Group | Stage 2, Group 2 Older Adults, ASP3772 Low Dose | Stage 2, Group 2 Older Adults, ASP3772 Medium Dose | Stage 2, Group 2 Older Adults, ASP3772 High Dose
Number analyzed (Participants) | 98 | 106 | 86
ln(titers)
  Serotype 1, Day 30 | 8.3 [8.0 to 8.7] | 8.6 [8.3 to 8.9] | 8.7 [8.3 to 9.1]
  Serotype 2, Day 30 | 9.3 [9.0 to 9.6] | 9.4 [9.1 to 9.7] | 9.7 [9.4 to 10.0]
  Serotype 3, Day 30 | 6.8 [6.5 to 7.1] | 7.2 [6.9 to 7.5] | 7.4 [7.1 to 7.7]
  Serotype 4, Day 30 | 7.2 [6.8 to 7.5] | 7.4 [7.1 to 7.7] | 7.4 [7.1 to 7.8]
  Serotype 5, Day 30 | 8.2 [7.8 to 8.6] | 8.2 [7.8 to 8.6] | 8.6 [8.1 to 9.0]
  Serotype 6A, Day 30 | 8.0 [7.6 to 8.5] | 8.2 [7.8 to 8.6] | 8.4 [7.9 to 8.8]
  Serotype 6B, Day 30 | 8.1 [7.6 to 8.5] | 8.4 [8.0 to 8.8] | 8.7 [8.2 to 9.1]
  Serotype 7F, Day 30 | 8.4 [8.1 to 8.8] | 8.5 [8.2 to 8.8] | 8.5 [8.1 to 8.9]
  Serotype 8, Day 30 | 9.0 [8.8 to 9.3] | 9.1 [8.9 to 9.4] | 9.7 [9.4 to 10.0]
  Serotype 9N, Day 30 | 8.6 [8.2 to 8.9] | 8.7 [8.4 to 9.1] | 9.2 [8.9 to 9.6]
  Serotype 9V, Day 30 | 7.9 [7.6 to 8.3] | 8.2 [7.9 to 8.5] | 8.4 [8.1 to 8.8]
  Serotype 10A, Day 30 | 9.2 [8.8 to 9.6] | 9.4 [9.0 to 9.7] | 9.7 [9.3 to 10.1]
  Serotype 11A, Day 30 | 8.1 [7.8 to 8.4] | 8.2 [7.9 to 8.5] | 8.6 [8.2 to 8.9]
  Serotype 12F, Day 30 | 6.4 [5.9 to 6.9] | 6.6 [6.1 to 7.0] | 6.6 [6.1 to 7.1]
  Serotype 14, Day 30 | 8.8 [8.3 to 9.2] | 9.0 [8.6 to 9.4] | 9.3 [8.9 to 9.8]
  Serotype 15B, Day 30 | 9.1 [8.7 to 9.5] | 9.4 [9.1 to 9.7] | 10.0 [9.6 to 10.3]
  Serotype 17F, Day 30 | 9.0 [8.7 to 9.3] | 9.2 [8.9 to 9.5] | 9.4 [9.1 to 9.8]
  Serotype 18C, Day 30 | 8.0 [7.6 to 8.3] | 8.5 [8.2 to 8.9] | 8.5 [8.1 to 8.9]
  Serotype 19A, Day 30 | 8.8 [8.4 to 9.1] | 9.0 [8.7 to 9.4] | 9.1 [8.7 to 9.5]
  Serotype 19F, Day 30 | 8.5 [8.1 to 8.9] | 8.9 [8.5 to 9.2] | 9.1 [8.8 to 9.5]
  Serotype 20B, Day 30 | 6.9 [6.6 to 7.3] | 7.0 [6.7 to 7.4] | 7.4 [7.0 to 7.8]
  Serotype 22F, Day 30 | 8.1 [7.8 to 8.4] | 8.2 [7.9 to 8.5] | 8.6 [8.3 to 8.9]
  Serotype 23F, Day 30 | 7.8 [7.4 to 8.2] | 7.8 [7.4 to 8.1] | 8.1 [7.7 to 8.5]
  Serotype 33F, Day 30 | 9.5 [9.1 to 9.9] | 9.7 [9.4 to 10.1] | 9.7 [9.3 to 10.1]
Statistical Analysis 1: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 Medium Dose; Serotype 1, Day 30; Test type: Other; p = 0.213, ANCOVA; Mean Difference = 0.3, 95% CI 2-sided [-0.1 to 0.7]
Statistical Analysis 2: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 1, Day 30; Test type: Other; p = 0.097, ANCOVA; Mean Difference = 0.4, 95% CI 2-sided [-0.1 to 0.8]
Statistical Analysis 3: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 1, Day 30; Test type: Other; p = 0.631, ANCOVA; Mean Difference = 0.1, 95% CI 2-sided [-0.3 to 0.5]
Statistical Analysis 4: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 Medium Dose; Serotype 2, Day 30; Test type: Other; p = 0.699, ANCOVA; Mean Difference = 0.1, 95% CI 2-sided [-0.3 to 0.4]
Statistical Analysis 5: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 2, Day 30; Test type: Other; p = 0.042, ANCOVA; Mean Difference = 0.4, 95% CI 2-sided [0.0 to 0.7]
Statistical Analysis 6: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 2, Day 30; Test type: Other; p = 0.092, ANCOVA; Mean Difference = 0.3, 95% CI 2-sided [-0.1 to 0.7]
Statistical Analysis 7: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 Medium Dose; Serotype 3, Day 30; Test type: Other; p = 0.007, ANCOVA; Mean Difference = 0.5, 95% CI 2-sided [0.1 to 0.8]
Statistical Analysis 8: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 3, Day 30; Test type: Other; p < .001, ANCOVA; Mean Difference = 0.7, 95% CI 2-sided [0.3 to 1.0]
Statistical Analysis 9: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 3, Day 30; Test type: Other; p = 0.237, ANCOVA; Mean Difference = 0.2, 95% CI 2-sided [-0.1 to 0.6]
Statistical Analysis 10: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 Medium Dose; Serotype 4, Day 30; Test type: Other; p = 0.248, ANCOVA; Mean Difference = 0.2, 95% CI 2-sided [-0.2 to 0.6]
Statistical Analysis 11: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 4, Day 30; Test type: Other; p = 0.193, ANCOVA; Mean Difference = 0.3, 95% CI 2-sided [-0.1 to 0.7]
Statistical Analysis 12: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 4, Day 30; Test type: Other; p = 0.838, ANCOVA; Mean Difference = 0.0, 95% CI 2-sided [-0.4 to 0.5]
Statistical Analysis 13: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 Medium Dose; Serotype 5, Day 30; Test type: Other; p = 0.898, ANCOVA; Mean Difference = 0.0, 95% CI 2-sided [-0.5 to 0.4]
Statistical Analysis 14: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 5, Day 30; Test type: Other; p = 0.143, ANCOVA; Mean Difference = 0.4, 95% CI 2-sided [-0.1 to 0.9]
Statistical Analysis 15: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 5, Day 30; Test type: Other; p = 0.108, ANCOVA; Mean Difference = 0.4, 95% CI 2-sided [-0.1 to 0.9]
Statistical Analysis 16: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 Medium Dose; Serotype 6A, Day 30; Test type: Other; p = 0.396, ANCOVA; Mean Difference = 0.2, 95% CI 2-sided [-0.3 to 0.7]
Statistical Analysis 17: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 6A, Day 30; Test type: Other; p = 0.182, ANCOVA; Mean Difference = 0.3, 95% CI 2-sided [-0.2 to 0.9]
Statistical Analysis 18: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 6A, Day 30; Test type: Other; p = 0.593, ANCOVA; Mean Difference = 0.1, 95% CI 2-sided [-0.4 to 0.6]
Statistical Analysis 19: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 6B, Day 30; Test type: Other; p = 0.186, ANCOVA; Mean Difference = 0.4, 95% CI 2-sided [-0.2 to 0.9]
Statistical Analysis 20: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 6B, Day 30; Test type: Other; p = 0.038, ANCOVA; Mean Difference = 0.6, 95% CI 2-sided [0.0 to 1.1]
Statistical Analysis 21: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 6B, Day 30; Test type: Other; p = 0.408, ANCOVA; Mean Difference = 0.2, 95% CI 2-sided [-0.3 to 0.8]
Statistical Analysis 22: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 Medium Dose; Serotype 7F, Day 30; Test type: Other; p = 0.805, ANCOVA; Mean Difference = 0.1, 95% CI 2-sided [-0.3 to 0.4]
Statistical Analysis 23: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 7F, Day 30; Test type: Other; p = 0.711, ANCOVA; Mean Difference = 0.1, 95% CI 2-sided [-0.3 to 0.5]
Statistical Analysis 24: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 7F, Day 30; Test type: Other; p = 0.891, ANCOVA; Mean Difference = 0.0, 95% CI 2-sided [-0.4 to 0.4]
Statistical Analysis 25: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 Medium Dose; Serotype 8, Day 30; Test type: Other; p = 0.649, ANCOVA; Mean Difference = 0.1, 95% CI 2-sided [-0.3 to 0.4]
Statistical Analysis 26: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 8, Day 30; Test type: Other; p < .001, ANCOVA; Mean Difference = 0.7, 95% CI 2-sided [0.3 to 1.0]
Statistical Analysis 27: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 8, Day 30; Test type: Other; p < .001, ANCOVA; Mean Difference = 0.6, 95% CI 2-sided [0.3 to 0.9]
Statistical Analysis 28: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 Medium Dose; Serotype 9N, Day 30; Test type: Other; p = 0.454, ANCOVA; Mean Difference = 0.2, 95% CI 2-sided [-0.2 to 0.5]
Statistical Analysis 29: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 9N, Day 30; Test type: Other; p = 0.003, ANCOVA; Mean Difference = 0.6, 95% CI 2-sided [0.2 to 1.0]
Statistical Analysis 30: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 9N, Day 30; Test type: Other; p = 0.021, ANCOVA; Mean Difference = 0.5, 95% CI 2-sided [0.1 to 0.9]
Statistical Analysis 31: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 Medium Dose; Serotype 9V, Day 30; Test type: Other; p = 0.205, ANCOVA; Mean Difference = 0.3, 95% CI 2-sided [-0.1 to 0.6]
Statistical Analysis 32: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 9V, Day 30; Test type: Other; p = 0.015, ANCOVA; Mean Difference = 0.5, 95% CI 2-sided [0.1 to 0.9]
Statistical Analysis 33: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 9V, Day 30; Test type: Other; p = 0.209, ANCOVA; Mean Difference = 0.3, 95% CI 2-sided [-0.1 to 0.7]
Statistical Analysis 34: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 Medium Dose; Serotype 10A, Day 30; Test type: Other; p = 0.502, ANCOVA; Mean Difference = 0.2, 95% CI 2-sided [-0.3 to 0.6]
Statistical Analysis 35: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 10A, Day 30; Test type: Other; p = 0.054, ANCOVA; Mean Difference = 0.5, 95% CI 2-sided [0.0 to 1.0]
Statistical Analysis 36: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 10A, Day 30; Test type: Other; p = 0.190, ANCOVA; Mean Difference = 0.3, 95% CI 2-sided [-0.2 to 0.8]
Statistical Analysis 37: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 Medium Dose; Serotype 11A, Day 30; Test type: Other; p = 0.616, ANCOVA; Mean Difference = 0.1, 95% CI 2-sided [-0.3 to 0.4]
Statistical Analysis 38: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 11A, Day 30; Test type: Other; p = 0.018, ANCOVA; Mean Difference = 0.4, 95% CI 2-sided [0.1 to 0.8]
Statistical Analysis 39: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 11A, Day 30; Test type: Other; p = 0.056, ANCOVA; Mean Difference = 0.4, 95% CI 2-sided [0.0 to 0.7]
Statistical Analysis 40: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 Medium Dose; Serotype 12F, Day 30; Test type: Other; p = 0.527, ANCOVA; Mean Difference = 0.2, 95% CI 2-sided [-0.4 to 0.7]
Statistical Analysis 41: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 12F, Day 30; Test type: Other; p = 0.444, ANCOVA; Mean Difference = 0.2, 95% CI 2-sided [-0.4 to 0.8]
Statistical Analysis 42: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 12F, Day 30; Test type: Other; p = 0.869, ANCOVA; Mean Difference = 0.0, 95% CI 2-sided [-0.5 to 0.6]
Statistical Analysis 43: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 Medium Dose; Serotype 14, Day 30; Test type: Other; p = 0.305, ANCOVA; Mean Difference = 0.3, 95% CI 2-sided [-0.2 to 0.7]
Statistical Analysis 44: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 14, Day 30; Test type: Other; p = 0.046, ANCOVA; Mean Difference = 0.5, 95% CI 2-sided [0.0 to 1.0]
Statistical Analysis 45: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 14, Day 30; Test type: Other; p = 0.299, ANCOVA; Mean Difference = 0.3, 95% CI 2-sided [-0.2 to 0.8]
Statistical Analysis 46: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 Medium Dose; Serotype 15B, Day 30; Test type: Other; p = 0.140, ANCOVA; Mean Difference = 0.3, 95% CI 2-sided [-0.1 to 0.7]
Statistical Analysis 47: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 15B, Day 30; Test type: Other; p < .001, ANCOVA; Mean Difference = 0.9, 95% CI 2-sided [0.4 to 1.3]
Statistical Analysis 48: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 15B, Day 30; Test type: Other; p = 0.012, ANCOVA; Mean Difference = 0.6, 95% CI 2-sided [0.1 to 1.0]
Statistical Analysis 49: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 Medium Dose; Serotype 17F, Day 30; Test type: Other; p = 0.200, ANCOVA; Mean Difference = 0.2, 95% CI 2-sided [-0.1 to 0.6]
Statistical Analysis 50: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 17F, Day 30; Test type: Other; p = 0.037, ANCOVA; Mean Difference = 0.4, 95% CI 2-sided [0.0 to 0.8]
Statistical Analysis 51: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 17F, Day 30; Test type: Other; p = 0.380, ANCOVA; Mean Difference = 0.2, 95% CI 2-sided [-0.2 to 0.6]
Statistical Analysis 52: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 Medium Dose; Serotype 18C, Day 30; Test type: Other; p = 0.006, ANCOVA; Mean Difference = 0.6, 95% CI 2-sided [0.2 to 1.0]
Statistical Analysis 53: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 18C, Day 30; Test type: Other; p = 0.018, ANCOVA; Mean Difference = 0.5, 95% CI 2-sided [0.1 to 1.0]
Statistical Analysis 54: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 18C, Day 30; Test type: Other; p = 0.810, ANCOVA; Mean Difference = -0.1, 95% CI 2-sided [-0.5 to 0.4]
Statistical Analysis 55: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 Medium Dose; Serotype 19A, Day 30; Test type: Other; p = 0.173, ANCOVA; Mean Difference = 0.3, 95% CI 2-sided [-0.1 to 0.7]
Statistical Analysis 56: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 19A, Day 30; Test type: Other; p = 0.096, ANCOVA; Mean Difference = 0.4, 95% CI 2-sided [-0.1 to 0.8]
Statistical Analysis 57: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 19A, Day 30; Test type: Other; p = 0.710, ANCOVA; Mean Difference = 0.1, 95% CI 2-sided [-0.3 to 0.5]
Statistical Analysis 58: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 Medium Dose; Serotype 19F, Day 30; Test type: Other; p = 0.100, ANCOVA; Mean Difference = 0.4, 95% CI 2-sided [-0.1 to 0.8]
Statistical Analysis 59: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 19F, Day 30; Test type: Other; p = 0.007, ANCOVA; Mean Difference = 0.6, 95% CI 2-sided [0.2 to 1.1]
Statistical Analysis 60: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 19F, Day 30; Test type: Other; p = 0.251, ANCOVA; Mean Difference = 0.3, 95% CI 2-sided [-0.2 to 0.7]
Statistical Analysis 61: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 Medium Dose; Serotype 20B, Day 30; Test type: Other; p = 0.618, ANCOVA; Mean Difference = 0.1, 95% CI 2-sided [-0.3 to 0.5]
Statistical Analysis 62: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 20B, Day 30; Test type: Other; p = 0.041, ANCOVA; Mean Difference = 0.5, 95% CI 2-sided [0.0 to 0.9]
Statistical Analysis 63: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 20B, Day 30; Test type: Other; p = 0.111, ANCOVA; Mean Difference = 0.3, 95% CI 2-sided [-0.1 to 0.8]
Statistical Analysis 64: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 Medium Dose; Serotype 22F, Day 30; Test type: Other; p = 0.758, ANCOVA; Mean Difference = 0.1, 95% CI 2-sided [-0.3 to 0.4]
Statistical Analysis 65: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 22F, Day 30; Test type: Other; p = 0.012, ANCOVA; Mean Difference = 0.5, 95% CI 2-sided [0.1 to 0.9]
Statistical Analysis 66: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 22F, Day 30; Test type: Other; p = 0.025, ANCOVA; Mean Difference = 0.4, 95% CI 2-sided [0.1 to 0.8]
Statistical Analysis 67: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 Medium Dose; Serotype 23F, Day 30; Test type: Other; p = 0.912, ANCOVA; Mean Difference = 0.0, 95% CI 2-sided [-0.5 to 0.4]
Statistical Analysis 68: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 23F, Day 30; Test type: Other; p = 0.174, ANCOVA; Mean Difference = 0.3, 95% CI 2-sided [-0.1 to 0.8]
Statistical Analysis 69: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 23F, Day 30; Test type: Other; p = 0.138, ANCOVA; Mean Difference = 0.3, 95% CI 2-sided [-0.1 to 0.8]
Statistical Analysis 70: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 Medium Dose; Serotype 33F, Day 30; Test type: Other; p = 0.267, ANCOVA; Mean Difference = 0.2, 95% CI 2-sided [-0.2 to 0.7]
Statistical Analysis 71: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 33F, Day 30; Test type: Other; p = 0.300, ANCOVA; Mean Difference = 0.2, 95% CI 2-sided [-0.2 to 0.7]
Statistical Analysis 72: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 2 Older Adults, ASP3772 High Dose; Serotype 33F, Day 30; Test type: Other; p = 0.982, ANCOVA; Mean Difference = 0.0, 95% CI 2-sided [-0.4 to 0.4]

25. Secondary Outcome: GMTs for Unique Serotype OPA Titer [Stage 2, Group 2 and Group 3]
Description: as for outcome 18
Time Frame: At Day 30
Population: The analysis was performed on the Full Analysis Set which consisted of all randomized participants who received a vaccination in this study with either ASP3772 or PPSV23, had at least 1 post vaccination measurement and for whom immunogenicity data was collected for specific serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Stage 2, Group 2 Older Adults, ASP3772 Low Dose | Stage 2, Group 2 Older Adults, ASP3772 Medium Dose | Stage 2, Group 2 Older Adults, ASP3772 High Dose | Stage 2, Group 3, PPSV23 Comparator
Number analyzed (Participants) | 97 | 105 | 84 | 107
Titers
  Serotype 2: number analyzed (Participants) | 96 | 105 | 84 | 107
  Serotype 2 | 1506.6 [1217.8 to 1864.0] | 1323.6 [1064.8 to 1645.3] | 2130.1 [1720.8 to 2636.7] | 1012.3 [779.7 to 1314.2]
  Serotype 8: number analyzed (Participants) | 96 | 104 | 79 | 98
  Serotype 8 | 1297.6 [1039.3 to 1620.1] | 1310.5 [997.2 to 1722.4] | 2792.4 [2202.5 to 3540.3] | 1342.6 [1025.0 to 1758.7]
  Serotype 9N: number analyzed (Participants) | 97 | 100 | 80 | 103
  Serotype 9N | 3200.2 [2433.1 to 4209.3] | 3814.9 [3162.7 to 4601.6] | 5279.3 [4200.6 to 6635.0] | 2362.1 [1788.1 to 3120.3]
  Serotype 10A: number analyzed (Participants) | 97 | 102 | 80 | 102
  Serotype 10A | 1958.5 [1387.7 to 2764.1] | 2574.0 [1874.3 to 3535.0] | 2912.5 [1926.3 to 4403.4] | 898.1 [580.6 to 1389.4]
  Serotype 11A: number analyzed (Participants) | 96 | 102 | 81 | 104
  Serotype 11A | 427.5 [322.6 to 566.4] | 509.4 [400.6 to 647.7] | 872.7 [657.7 to 1158.0] | 359.5 [269.7 to 479.3]
  Serotype 12F: number analyzed (Participants) | 95 | 102 | 82 | 95
  Serotype 12F | 1364.7 [972.2 to 1915.7] | 1014.9 [730.3 to 1410.5] | 1712.0 [1185.4 to 2472.4] | 1133.9 [775.0 to 1658.9]
  Serotype 15B: number analyzed (Participants) | 88 | 86 | 72 | 102
  Serotype 15B | 6095.8 [4420.5 to 8406.1] | 4539.1 [3479.4 to 5921.4] | 6988.4 [5235.6 to 9328.0] | 4147.3 [3039.9 to 5658.3]
  Serotype 17F: number analyzed (Participants) | 97 | 103 | 81 | 106
  Serotype 17F | 4308.7 [3335.3 to 5566.2] | 3528.6 [2820.2 to 4414.9] | 5567.0 [4337.9 to 7144.3] | 1653.4 [1154.7 to 2367.5]
  Serotype 20B: number analyzed (Participants) | 92 | 95 | 73 | 104
  Serotype 20B | 15461.3 [11110.3 to 21516.4] | 12442.1 [9136.1 to 16944.4] | 23411.3 [16037.8 to 34174.7] | 1708.7 [1215.2 to 2402.7]
  Serotype 22F: number analyzed (Participants) | 93 | 93 | 81 | 96
  Serotype 22F | 2017.5 [1479.5 to 2751.2] | 1741.4 [1331.9 to 2276.9] | 2442.6 [1888.6 to 3159.0] | 1126.2 [759.6 to 1669.9]
  Serotype 33F: number analyzed (Participants) | 95 | 101 | 83 | 106
  Serotype 33F | 6822.7 [4904.1 to 9491.9] | 6265.0 [4847.4 to 8097.3] | 8579.4 [6421.0 to 11463.2] | 5072.8 [3729.5 to 6900.0]
Statistical Analysis 1: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 2; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.49, 95% CI 2-sided [1.06 to 2.08]
Statistical Analysis 2: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 8; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.97, 95% CI 2-sided [0.68 to 1.37]
Statistical Analysis 3: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 9N; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.35, 95% CI 2-sided [0.92 to 2.00]
Statistical Analysis 4: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 10A; Test type: Other; t-test, 2 sided; Ratio of GMT = 2.18, 95% CI 2-sided [1.25 to 3.79]
Statistical Analysis 5: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 11A; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.19, 95% CI 2-sided [0.80 to 1.77]
Statistical Analysis 6: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 12F; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.20, 95% CI 2-sided [0.73 to 2.00]
Statistical Analysis 7: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 15B; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.47, 95% CI 2-sided [0.94 to 2.29]
Statistical Analysis 8: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 17F; Test type: Other; t-test, 2 sided; Ratio of GMT = 2.61, 95% CI 2-sided [1.68 to 4.04]
Statistical Analysis 9: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 20B; Test type: Other; t-test, 2 sided; Ratio of GMT = 9.05, 95% CI 2-sided [5.65 to 14.50]
Statistical Analysis 10: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 22F; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.79, 95% CI 2-sided [1.09 to 2.95]
Statistical Analysis 11: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 3, PPSV23 Comparator; Test type: Other — Serotype 33F; t-test, 2 sided; Ratio of GMT = 1.34, 95% CI 2-sided [0.86 to 2.11]
Statistical Analysis 12: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 2; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.31, 95% CI 2-sided [0.93 to 1.83]
Statistical Analysis 13: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 8; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.98, 95% CI 2-sided [0.67 to 1.43]
Statistical Analysis 14: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 9N; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.62, 95% CI 2-sided [1.62 to 2.26]
Statistical Analysis 15: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 10A; Test type: Other; t-test, 2 sided; Ratio of GMT = 2.87, 95% CI 2-sided [1.68 to 4.90]
Statistical Analysis 16: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 11A; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.42, 95% CI 2-sided [0.98 to 2.06]
Statistical Analysis 17: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 12F; Test type: Other; t-test, 2 sided; Ratio of GMT = 0.90, 95% CI 2-sided [0.54 to 1.48]
Statistical Analysis 18: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 15B; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.09, 95% CI 2-sided [0.73 to 1.64]
Statistical Analysis 19: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 17F; Test type: Other; t-test, 2 sided; Ratio of GMT = 2.13, 95% CI 2-sided [1.40 to 3.25]
Statistical Analysis 20: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 20B; Test type: Other; t-test, 2 sided; Ratio of GMT = 7.28, 95% CI 2-sided [4.61 to 11.50]
Statistical Analysis 21: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 22F; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.55, 95% CI 2-sided [0.96 to 2.48]
Statistical Analysis 22: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 33F; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.24, 95% CI 2-sided [0.83 to 1.84]
Statistical Analysis 23: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 2; Test type: Other; t-test, 2 sided; Ratio of GMT = 2.10, 95% CI 2-sided [1.51 to 2.94]
Statistical Analysis 24: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 8; Test type: Other; t-test, 2 sided; Ratio of GMT = 2.08, 95% CI 2-sided [1.46 to 2.97]
Statistical Analysis 25: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 9N; Test type: Other; t-test, 2 sided; Ratio of GMT = 2.24, 95% CI 2-sided [1.56 to 3.20]
Statistical Analysis 26: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 10A; Test type: Other; t-test, 2 sided; Ratio of GMT = 3.24, 95% CI 2-sided [1.79 to 5.89]
Statistical Analysis 27: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 11A; Test type: Other; t-test, 2 sided; Ratio of GMT = 2.43, 95% CI 2-sided [1.63 to 3.62]
Statistical Analysis 28: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 12 F; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.51, 95% CI 2-sided [0.89 to 2.55]
Statistical Analysis 29: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 15B; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.69, 95% CI 2-sided [1.11 to 2.57]
Statistical Analysis 30: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 17F; Test type: Other; t-test, 2 sided; Ratio of GMT = 3.37, 95% CI 2-sided [2.18 to 5.20]
Statistical Analysis 31: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 20B; Test type: Other; t-test, 2 sided; Ratio of GMT = 13.70, 95% CI 2-sided [8.26 to 22.72]
Statistical Analysis 32: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 22F; Test type: Other; t-test, 2 sided; Ratio of GMT = 2.17, 95% CI 2-sided [1.36 to 3.46]
Statistical Analysis 33: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 33F; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.69, 95% CI 2-sided [1.11 to 2.57]

26. Secondary Outcome: GMCs for Unique Serotypes IgG, [Stage 2, Group 2 and Group 3]
Description: Immunogenicity was measured in terms of IgG GMCs and expressed as titers. The assessed serotypes were: 2, 8, 9N, 10A, 11A, 12F, 15B, 17F, 20B, 22F, 33F.
Time Frame: At Day 30
Population: The analysis was performed on the FAS which consisted of all enrolled participants in Stage 2, Group 3 who received a vaccination in this study with PPSV23 and had at least 1 post vaccination measurement.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Stage 2, Group 2 Older Adults, ASP3772 Low Dose | Stage 2, Group 2 Older Adults, ASP3772 Medium Dose | Stage 2, Group 2 Older Adults, ASP3772 High Dose | Stage 2, Group 3, PPSV23 Comparator
Number analyzed (Participants) | 98 | 106 | 86 | 110
Titers
  Serotype 2: number analyzed (Participants) | 98 | 106 | 86 | 108
  Serotype 2 | 12372.5 [9734.3 to 15725.7] | 13002.6 [9984.9 to 16932.5] | 18046.8 [14062.8 to 23159.5] | 9152.0 [6999.2 to 11966.8]
  Serotype 8: number analyzed (Participants) | 98 | 106 | 86 | 108
  Serotype 8 | 9677.9 [7671.1 to 12209.7] | 10169.1 [7940.9 to 13022.6] | 19090.8 [15224.8 to 23938.5] | 6416.8 [4968.2 to 8287.6]
  Serotype 9N: number analyzed (Participants) | 98 | 106 | 86 | 108
  Serotype 9N | 5768.2 [4408.9 to 7546.6] | 6616.2 [4919.6 to 8897.8] | 10826.9 [8103.3 to 14465.7] | 3619.7 [2761.6 to 4744.5]
  Serotype 10A: number analyzed (Participants) | 98 | 106 | 86 | 108
  Serotype 10A | 10809.8 [7891.5 to 14807.3] | 12474.3 [8946.9 to 17392.2] | 17483.9 [12026.3 to 25418.2] | 4815.5 [3557.3 to 6518.8]
  Serotype 11A: number analyzed (Participants) | 98 | 106 | 86 | 108
  Serotype 11A | 4445.2 [3442.1 to 5740.5] | 4602.5 [3584.5 to 5909.6] | 6928.5 [5266.2 to 9115.4] | 2423.4 [1857.6 to 3161.4]
  Serotype 12F: number analyzed (Participants) | 98 | 106 | 86 | 108
  Serotype 12F | 556.1 [382.8 to 808.0] | 675.3 [462.1 to 986.8] | 696.8 [441.3 to 1100.1] | 424.4 [290.2 to 620.5]
  Serotype 15B: number analyzed (Participants) | 98 | 106 | 86 | 108
  Serotype 15B | 9320.5 [6869.4 to 12646.0] | 12611.9 [9628.3 to 16520.1] | 22041.9 [15842.8 to 30666.5] | 7515.1 [5496.3 to 10275.5]
  Serotype 17F: number analyzed (Participants) | 98 | 106 | 86 | 108
  Serotype 17F | 9259.1 [6977.1 to 12287.6] | 11508.5 [9042.1 to 14647.5] | 14067.7 [10377.3 to 19070.6] | 3517.3 [2520.6 to 4908.1]
  Serotype 20B: number analyzed (Participants) | 98 | 106 | 86 | 108
  Serotype 20B | 863.3 [646.3 to 1153.1] | 991.4 [741.0 to 1326.5] | 1355.5 [979.5 to 1875.8] | 355.3 [264.0 to 478.2]
  Serotype 22F: number analyzed (Participants) | 98 | 106 | 86 | 108
  Serotype 22F | 3385.1 [2624.9 to 4365.5] | 3577.6 [2755.1 to 4645.6] | 5462.2 [4218.3 to 7072.9] | 1359.0 [1018.7 to 1813.1]
  Serotype 33F: number analyzed (Participants) | 98 | 106 | 86 | 108
  Serotype 33F | 15822.1 [11471.2 to 21823.3] | 19432.8 [14796.7 to 25521.3] | 19959.6 [14321.7 to 27817.0] | 9459.6 [7222.2 to 12390.2]
Statistical Analysis 1: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 2; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.35, 95% CI 2-sided [0.95 to 1.93]
Statistical Analysis 2: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 8; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.51, 95% CI 2-sided [1.07 to 2.13]
Statistical Analysis 3: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 9N; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.59, 95% CI 2-sided [1.09 to 2.33]
Statistical Analysis 4: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 10A; Test type: Other; t-test, 2 sided; Ratio of GMT = 2.24, 95% CI 2-sided [1.45 to 3.47]
Statistical Analysis 5: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 11A; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.83, 95% CI 2-sided [1.27 to 2.65]
Statistical Analysis 6: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 12F; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.31, 95% CI 2-sided [0.77 to 2.23]
Statistical Analysis 7: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 15B; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.24, 95% CI 2-sided [0.80 to 1.91]
Statistical Analysis 8: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 17F; Test type: Other; t-test, 2 sided; Ratio of GMT = 2.63, 95% CI 2-sided [1.70 to 4.07]
Statistical Analysis 9: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 20B; Test type: Other; t-test, 2 sided; Ratio of GMT = 2.43, 95% CI 2-sided [1.61 to 3.67]
Statistical Analysis 10: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 22F; Test type: Other; t-test, 2 sided; Ratio of GMT = 2.49, 95% CI 2-sided [1.70 to 3.65]
Statistical Analysis 11: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Low Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 33F; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.67, 95% CI 2-sided [1.10 to 2.54]
Statistical Analysis 12: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 2; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.42, 95% CI 2-sided [0.98 to 2.07]
Statistical Analysis 13: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 8; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.58, 95% CI 2-sided [1.11 to 2.26]
Statistical Analysis 14: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 9N; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.83, 95% CI 2-sided [1.23 to 2.72]
Statistical Analysis 15: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 10A; Test type: Other; Ratio of GMT = 2.59, 95% CI 2-sided [1.66 to 4.05]
Statistical Analysis 16: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 11A; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.90, 95% CI 2-sided [1.32 to 2.73]
Statistical Analysis 17: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 12F; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.59, 95% CI 2-sided [0.93 to 2.71]
Statistical Analysis 18: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 15B; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.68, 95% CI 2-sided [1.11 to 2.53]
Statistical Analysis 19: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 17F; Test type: Other; t-test, 2 sided; Ratio of GMT = 3.27, 95% CI 2-sided [2.17 to 4.93]
Statistical Analysis 20: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 20B; Test type: Other; t-test, 2 sided; Ratio of GMT = 2.79, 95% CI 2-sided [1.85 to 4.22]
Statistical Analysis 21: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 22F; Test type: Other; t-test, 2 sided; Ratio of GMT = 2.63, 95% CI 2-sided [1.79 to 3.88]
Statistical Analysis 22: Comparison: Stage 2, Group 2 Older Adults, ASP3772 Medium Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 33F; Test type: Other; t-test, 2 sided; Ratio of GMT = 2.05, 95% CI 2-sided [1.40 to 3.01]
Statistical Analysis 23: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 2; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.97, 95% CI 2-sided [1.37 to 2.84]
Statistical Analysis 24: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 8; Test type: Other; t-test, 2 sided; Ratio of GMT = 2.98, 95% CI 2-sided [2.12 to 4.18]
Statistical Analysis 25: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 9N; Test type: Other; t-test, 2 sided; Ratio of GMT = 2.99, 95% CI 2-sided [2.02 to 4.44]
Statistical Analysis 26: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 10A; Test type: Other; t-test, 2 sided; Ratio of GMT = 3.63, 95% CI 2-sided [2.25 to 5.86]
Statistical Analysis 27: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 11A; Test type: Other; t-test, 2 sided; Ratio of GMT = 2.86, 95% CI 2-sided [1.96 to 4.18]
Statistical Analysis 28: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 12F; Test type: Other; t-test, 2 sided; Ratio of GMT = 1.64, 95% CI 2-sided [0.91 to 2.96]
Statistical Analysis 29: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 15B; Test type: Other; t-test, 2 sided; Ratio of GMT = 2.93, 95% CI 2-sided [1.87 to 4.61]
Statistical Analysis 30: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 17F; Test type: Other; t-test, 2 sided; Ratio of GMT = 4.00, 95% CI 2-sided [2.55 to 6.26]
Statistical Analysis 31: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 22F; Test type: Other; t-test, 2 sided; Ratio of GMT = 3.82, 95% CI 2-sided [2.46 to 5.91]
Statistical Analysis 32: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 22F; Test type: Other; t-test, 2 sided; Ratio of GMT = 4.02, 95% CI 2-sided [2.74 to 5.90]
Statistical Analysis 33: Comparison: Stage 2, Group 2 Older Adults, ASP3772 High Dose vs Stage 2, Group 3, PPSV23 Comparator; Serotype 33F; Test type: Other; t-test, 2 sided; Ratio of GMT = 2.11, 95% CI 2-sided [1.38 to 3.23]

ADVERSE EVENTS:
Time Frame: SAEs were collected from Day 1 to Day 180 (study end). Non-serious adverse events collected during 7 days post vaccination.
Description: The analysis was performed on the Safety Analysis Set (SAF) which consisted of all randomized participants who received a vaccination in this study with either ASP3772, PCV13 and PPSV23.
  Note: for Other Adverse Events Tenderness and Pain solicited events are mapped to 'Injection site pain' as Preferred Term. Hence if the same subject experiences at least once both Tenderness and Pain, he/she will count only once in n.
Arm/Group | Stage 1, Group 1 Adults, ASP3772 Low Dose | Stage 1, Group 1 Adults, ASP3772 Medium Dose | Stage 1, Group 1 Adults, ASP3772 High Dose | Stage 1, Group 1, PCV13 Pooled Comparator | Stage 2, Group 2 Older Adults, ASP3772 Low Dose | Stage 2, Group 2 Older Adults, ASP3772 Medium Dose | Stage 2, Group 2 Older Adults, ASP3772 High Dose | Stage 2, Group 2, PCV13 Pooled Comparator | Stage 2, Group 3, PPSV23 Comparator
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/31 | 0/32 | 0/33 | 0/100 | 1/107 | 0/86 | 0/97 | 0/113
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/31 | 0/32 | 0/33 | 4/100 | 5/107 | 1/86 | 0/97 | 0/113
Other Adverse Events (participants affected / at risk) | 22/30 | 24/31 | 28/32 | 29/33 | 56/100 | 68/107 | 65/86 | 56/97 | 4/113
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage 1, Group 1 Adults, ASP3772 Low Dose (N=30) | Stage 1, Group 1 Adults, ASP3772 Medium Dose (N=31) | Stage 1, Group 1 Adults, ASP3772 High Dose (N=32) | Stage 1, Group 1, PCV13 Pooled Comparator (N=33) | Stage 2, Group 2 Older Adults, ASP3772 Low Dose (N=100) | Stage 2, Group 2 Older Adults, ASP3772 Medium Dose (N=107) | Stage 2, Group 2 Older Adults, ASP3772 High Dose (N=86) | Stage 2, Group 2, PCV13 Pooled Comparator (N=97) | Stage 2, Group 3, PPSV23 Comparator (N=113)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestine adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal claudication (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage 1, Group 1 Adults, ASP3772 Low Dose (N=30) | Stage 1, Group 1 Adults, ASP3772 Medium Dose (N=31) | Stage 1, Group 1 Adults, ASP3772 High Dose (N=32) | Stage 1, Group 1, PCV13 Pooled Comparator (N=33) | Stage 2, Group 2 Older Adults, ASP3772 Low Dose (N=100) | Stage 2, Group 2 Older Adults, ASP3772 Medium Dose (N=107) | Stage 2, Group 2 Older Adults, ASP3772 High Dose (N=86) | Stage 2, Group 2, PCV13 Pooled Comparator (N=97) | Stage 2, Group 3, PPSV23 Comparator (N=113)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 7 (7) | 11 (11) | 13 (13) | 11 (11) | 26 (26) | 27 (27) | 17 (17) | 0 (0)
Headache (Nervous system disorders) | 6 (6) | 6 (6) | 7 (7) | 13 (14) | 13 (13) | 13 (13) | 10 (10) | 10 (10) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 2 (2) | 4 (4) | 6 (6) | 4 (4) | 15 (16) | 13 (13) | 6 (6) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 10 (10) | 13 (13) | 8 (8) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 6 (6) | 9 (9) | 5 (5) | 1 (1)
Fatigue (General disorders) | 7 (7) | 8 (8) | 10 (10) | 13 (13) | 18 (18) | 18 (18) | 22 (22) | 21 (21) | 1 (1)
Injection site erythema (General disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 4 (4) | 4 (4) | 6 (6) | 4 (4) | 1 (1)
Injection site induration (General disorders) | 0 (0) | 2 (2) | 1 (1) | 4 (4) | 2 (2) | 6 (6) | 4 (4) | 2 (2) | 0 (0)
Injection site pain (General disorders) | 17 (21) | 24 (26) | 25 (28) | 27 (34) | 41 (47) | 58 (61) | 53 (62) | 46 (52) | 1 (1)
Injection site swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 6 (6) | 4 (4) | 4 (4) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-12-04): https://cdn.clinicaltrials.gov/large-docs/02/NCT03803202/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-30): https://cdn.clinicaltrials.gov/large-docs/02/NCT03803202/SAP_001.pdf